CLINICAL TRIAL: NCT00023595
Title: Surgical Treatment for Ischemic Heart Failure (STICH)
Brief Title: Comparison of Surgical and Medical Treatment for Congestive Heart Failure and Coronary Artery Disease
Acronym: STICH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00018940; U01HL069009 (NIH); U01HL069010 (NIH); U01HL069011 (NIH); U01HL069012 (NIH); U01HL069013 (NIH); U01HL069015 (NIH); U01HL072683 (NIH); R01HL105853 (NIH); Pro00010463 (Other: Duke IRB)
Record Dates: First submitted 2001-09-11; First posted 2001-09-11 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Failure, Congestive; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Failure; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- H01: Medication (Active Comparator): Medical therapy alone to treat Coronary Artery Disease
  Interventions: Drug: Active Medication Alone
- H01: Medication + CABG (Active Comparator): Coronary artery bypass graft surgery (CABG) plus Medication to treat coronary artery disease
  Interventions: Procedure: CABG surgery plus MED
- H02: Medication+CABG (Active Comparator): Coronary artery bypass graft surgery (CABG) plus Medication to treat coronary artery disease
  Interventions: Procedure: CABG surgery plus MED
- H02: Medication+CABG+SVR (Active Comparator): CABG plus Medication and Surgical ventricular reconstruction (SVR)
  Interventions: Procedure: CABG plus MED and SVR

INTERVENTIONS:
Procedure: CABG surgery plus MED — CABG plus standard medication management for Coronary Artery Disease
  Arms: H01: Medication + CABG; H02: Medication+CABG
Drug: Active Medication Alone — Standard medication for coronary artery disease and heart failure management.
  Other Names: Standard medications for management of CAD and heart failure
  Arms: H01: Medication
Procedure: CABG plus MED and SVR — H02: the experimental arm receives active medical therapy and CABG and surgical ventricular restoration whereas the control group receives active medical therapy and CABG; for H01: the experimental arm receives active medical therapy and CABG whereas the control group receives active medical therapy alone
  Arms: H02: Medication+CABG+SVR

SUMMARY:
This study will compare medical therapy with coronary bypass surgery and/or surgical ventricular reconstruction for patients with congestive heart failure and coronary artery disease (CAD).

DETAILED DESCRIPTION:
BACKGROUND:

Congestive heart failure afflicts approximately five million Americans and is the leading cause of hospitalization in Americans over the age of 65. Most cases of congestive heart failure are due to CAD. Surprisingly little is known about the relative benefits of medical versus surgical therapy for patients with obstructive coronary disease and congestive heart failure. Randomized studies of medical therapy versus bypass surgery for obstructive coronary disease were conducted in the 1970s and did not include the systematic use of aspirin, arterial conduits, or lipid-lowering medications. In addition, patients with ejection fractions below 35% were specifically excluded from the three large randomized studies of medical therapy versus bypass surgery. While observational data from the 1970s and early 1980s suggest a survival advantage associated with bypass surgery in patients with low ejection fraction and congestive heart failure, biases favoring the referral of the fittest of such patients for bypass surgery may have confounded these comparisons. In addition, medical therapy for congestive heart failure has improved dramatically over the past two decades. Thus, the choice of medical therapy versus bypass surgery for patients with congestive heart failure and obstructive coronary disease is usually decided by guesswork. This study is designed to provide a solid answer.

PURPOSE:

STICH is a multicenter, international, randomized trial that addresses two specific primary hypotheses in patients with clinical heart failure (HF) and left ventricular (LV) dysfunction who have coronary artery disease amenable to surgical revascularization.

The first hypothesis is that restoration of blood flow by means of coronary revascularization recovers chronic LV dysfunction and improves survival, as compared to intensive medical therapy alone. The second hypothesis is that surgical ventricular restoration (SVR) to a more normal LV size improves survival free of subsequent hospitalization for cardiac cause compared to CABG alone.

Patients eligible for either medical therapy or CABG, but not eligible for the SVR procedure (Stratum A), will be randomized in equal proportions to medical therapy alone versus CABG plus medical therapy. Patients eligible for all three therapies (Stratum B) will be randomized in equal proportions to medical therapy alone, CABG plus medical therapy, and CABG plus SVR plus medical therapy. Patients whose severity of angina or CAD makes them inappropriate for medical therapy alone (Stratum C) will be randomized in equal proportions to CABG plus medical therapy versus CABG plus SVR plus medical therapy.

The overall target was to recruit 1200 patients into Hypothesis One and 1,000 patients into Hypothesis Two. Secondary endpoints include the role of myocardial viability, morbidity, economics, and quality of life. Core laboratories for quality of life/economics, cardiac magnetic resonance (CMR), echocardiography (ECHO), neurohormonal/cytokine/genetic (NCG), and radionuclide (RN) studies ensure consistent testing practices and standardization of data necessary to identify eligible patients and to address specific questions related to the stated hypotheses.

IMPORTANCE OF RESEARCH:

The most common cause of HF is no longer hypertension or valvular heart disease as it was in previous decades, but rather CAD. HF is a common worldwide disease and CAD is a frequent cause of HF initiation and progression. HF is responsible for approximately 1 million hospitalizations and 300,000 fatalities annually. The prevalence of HF is increasing, largely due to enhanced survival following acute myocardial infarction and other manifestations of CAD. No randomized trial has ever compared directly the long-term benefits of surgical, medical, or combined surgical and medical treatment of patients with ischemic HF. The STICH trial is the first trial to compare the long term benefits of surgical and medical treatment in patients with ischemic HF. Although modern medical therapy for HF modestly improves quality of life, a more aggressive approach with the surgical therapies being studied in the STICH trial may produce even greater improvements. The common clinical practice of not offering CABG to patients with LV dysfunction in regions found to be nonviable on noninvasive studies is not evidence-based. Since only those patients for whom intensive medical therapy is the only reasonable therapeutic alternative are excluded from this study, the results of the STICH trial should be applicable to most patients with CAD, HF, and systolic LV dysfunction. The results of the STICH trial will also establish whether measurements of neurohormonal and cytokine levels and genetic profiling are useful for directing patient management decisions, for monitoring the effectiveness of therapy, and for refining the optimal approach for selecting the treatment strategy most likely to be effective for the many of these patients.

ELIGIBILITY:
Inclusion Criteria:

* LV less than 35%, as defined by echocardiogram, left ventriculogram, CMR, or gated single photon emission computed tomography (SPECT) studies
* Coronary anatomy suitable for revascularization

Exclusion Criteria:

* Failure to provide informed consent.
* Aortic valvular heart disease clearly indicating the need for aortic valve repair or replacement.
* Cardiogenic shock (within 72 hours of randomization), as defined by the need for intraaortic balloon support or the requirement for intravenous inotropic support.
* Plan for percutaneous intervention of CAD.
* Recent acute MI judged to be an important cause of left ventricular dysfunction.
* History of more than 1 prior coronary bypass operation.
* Noncardiac illness with a life expectancy of less than 3 years.
* Noncardiac illness imposing substantial operative mortality.
* Conditions/circumstances likely to lead to poor treatment adherence (eg, history of poor compliance, alcohol or drug dependency, psychiatric illness, no fixed abode).
* Previous heart, kidney, liver, or lung transplantation.
* Current participation in another clinical trial in which a patient is taking an investigational drug or receiving an investigational medical device.

MED Therapy Eligibility Criteria

* Absence of left main CAD as defined by an intraluminal stenosis of 50% or greater.
* Absence of CCS III angina or greater (angina markedly limiting ordinary activity).

SVR Eligibility Criterion

• Dominant akinesia or dyskinesia of the anterior left ventricular wall amenable to SVR.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2136 (Actual)
Dates: Start 2002-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bonow, Principal Investigator — Radionuclide Core Lab, Northwestern University; Arthur Feldman, Principal Investigator — Neurohormonal Core Lab, Jefferson University; Eric Velazquez, MD, Principal Investigator — Clinical Coordinating Center, Duke University; Kerry Lee, Principal Investigator — Data Coordinating Center, Duke University; Daniel Mark, Principal Investigator — Economics and Quality of Life Core Lab, Duke University; Jae Oh, Principal Investigator — Echocardiographic Core Lab, Mayo Clinic; Gerald Pohost, Principal Investigator — Magnetic Resonance Imaging Core Lab, University of Southern California; Jean Rouleau, Study Chair — Université de Montréal; Julio A Panza, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Velazquez EJ, Lee KL, O'Connor CM, Oh JK, Bonow RO, Pohost GM, Feldman AM, Mark DB, Panza JA, Sopko G, Rouleau JL, Jones RH; STICH Investigators. The rationale and design of the Surgical Treatment for Ischemic Heart Failure (STICH) trial. J Thorac Cardiovasc Surg. 2007 Dec;134(6):1540-7. doi: 10.1016/j.jtcvs.2007.05.069. PMID 18023680
- [Derived] Wen B, Lu Y, Huang X, Du X, Sun F, Xie F, Liu C, Wang D. Influence and risk factors of postoperative infection after surgery for ischemic cardiomyopathy. Front Cardiovasc Med. 2023 Aug 24;10:1231556. doi: 10.3389/fcvm.2023.1231556. eCollection 2023. PMID 37692042
- [Derived] Ezad SM, Ryan M, Perera D. Can Percutaneous Coronary Intervention Revive a Failing Heart? Heart Int. 2022 Dec 21;16(2):72-74. doi: 10.17925/HI.2022.16.2.72. eCollection 2022. PMID 36741102
- [Derived] Chew DS, Cowper PA, Al-Khalidi H, Anstrom KJ, Daniels MR, Davidson-Ray L, Li Y, Michler RE, Panza JA, Pina IL, Rouleau JL, Velazquez EJ, Mark DB; STICH Investigators. Cost-Effectiveness of Coronary Artery Bypass Surgery Versus Medicine in Ischemic Cardiomyopathy: The STICH Randomized Clinical Trial. Circulation. 2022 Mar 15;145(11):819-828. doi: 10.1161/CIRCULATIONAHA.121.056276. Epub 2022 Jan 19. PMID 35044802
- [Derived] Farsky PS, White J, Al-Khalidi HR, Sueta CA, Rouleau JL, Panza JA, Velazquez EJ, O'Connor CM; Working Group and Surgical Treatment for Ischemic Heart Failure Trial Investigators. Optimal medical therapy with or without surgical revascularization and long-term outcomes in ischemic cardiomyopathy. J Thorac Cardiovasc Surg. 2022 Dec;164(6):1890-1899.e4. doi: 10.1016/j.jtcvs.2020.12.094. Epub 2021 Jan 7. PMID 33610365
- [Derived] Perry AS, Mann DL, Brown DL. Improvement of ejection fraction and mortality in ischaemic heart failure. Heart. 2020 Aug 25:heartjnl-2020-316975. doi: 10.1136/heartjnl-2020-316975. Online ahead of print. PMID 32843496
- [Derived] Howlett JG, Stebbins A, Petrie MC, Jhund PS, Castelvecchio S, Cherniavsky A, Sueta CA, Roy A, Pina IL, Wurm R, Drazner MH, Andersson B, Batlle C, Senni M, Chrzanowski L, Merkely B, Carson P, Desvigne-Nickens PM, Lee KL, Velazquez EJ, Al-Khalidi HR; STICH Trial Investigators. CABG Improves Outcomes in Patients With Ischemic Cardiomyopathy: 10-Year Follow-Up of the STICH Trial. JACC Heart Fail. 2019 Oct;7(10):878-887. doi: 10.1016/j.jchf.2019.04.018. Epub 2019 Sep 11. PMID 31521682
- [Derived] Panza JA, Ellis AM, Al-Khalidi HR, Holly TA, Berman DS, Oh JK, Pohost GM, Sopko G, Chrzanowski L, Mark DB, Kukulski T, Favaloro LE, Maurer G, Farsky PS, Tan RS, Asch FM, Velazquez EJ, Rouleau JL, Lee KL, Bonow RO. Myocardial Viability and Long-Term Outcomes in Ischemic Cardiomyopathy. N Engl J Med. 2019 Aug 22;381(8):739-748. doi: 10.1056/NEJMoa1807365. PMID 31433921
- [Derived] Nicolau JC, Stevens SR, Al-Khalidi HR, Jatene FB, Furtado RHM, Dallan LAO, Lisboa LAF, Desvigne-Nickens P, Haddad H, Jolicoeur EM, Petrie MC, Doenst T, Michler RE, Ohman EM, Maddury J, Ali I, Deja MA, Rouleau JL, Velazquez EJ, Hill JA. Does prior coronary angioplasty affect outcomes of surgical coronary revascularization? Insights from the STICH trial. Int J Cardiol. 2019 Sep 15;291:36-41. doi: 10.1016/j.ijcard.2019.03.029. Epub 2019 Mar 15. PMID 30929973
- [Derived] Ambrosy AP, Stevens SR, Al-Khalidi HR, Rouleau JL, Bouabdallaoui N, Carson PE, Adlbrecht C, Cleland JGF, Dabrowski R, Golba KS, Pina IL, Sueta CA, Roy A, Sopko G, Bonow RO, Velazquez EJ; STICH Trial Investigators. Burden of medical co-morbidities and benefit from surgical revascularization in patients with ischaemic cardiomyopathy. Eur J Heart Fail. 2019 Mar;21(3):373-381. doi: 10.1002/ejhf.1404. Epub 2019 Jan 30. PMID 30698316
- [Derived] Pellikka PA, She L, Holly TA, Lin G, Varadarajan P, Pai RG, Bonow RO, Pohost GM, Panza JA, Berman DS, Prior DL, Asch FM, Borges-Neto S, Grayburn P, Al-Khalidi HR, Miszalski-Jamka K, Desvigne-Nickens P, Lee KL, Velazquez EJ, Oh JK. Variability in Ejection Fraction Measured By Echocardiography, Gated Single-Photon Emission Computed Tomography, and Cardiac Magnetic Resonance in Patients With Coronary Artery Disease and Left Ventricular Dysfunction. JAMA Netw Open. 2018 Aug 3;1(4):e181456. doi: 10.1001/jamanetworkopen.2018.1456. PMID 30646130
- [Derived] Bouabdallaoui N, Stevens SR, Doenst T, Petrie MC, Al-Attar N, Ali IS, Ambrosy AP, Barton AK, Cartier R, Cherniavsky A, Demondion P, Desvigne-Nickens P, Favaloro RR, Gradinac S, Heinisch P, Jain A, Jasinski M, Jouan J, Kalil RAK, Menicanti L, Michler RE, Rao V, Smith PK, Zembala M, Velazquez EJ, Al-Khalidi HR, Rouleau JL; STICH Trial Investigators. Society of Thoracic Surgeons Risk Score and EuroSCORE-2 Appropriately Assess 30-Day Postoperative Mortality in the STICH Trial and a Contemporary Cohort of Patients With Left Ventricular Dysfunction Undergoing Surgical Revascularization. Circ Heart Fail. 2018 Nov;11(11):e005531. doi: 10.1161/CIRCHEARTFAILURE.118.005531. PMID 30571194
- [Derived] Andersson B, She L, Tan RS, Jeemon P, Mokrzycki K, Siepe M, Romanov A, Favaloro LE, Djokovic LT, Raju PK, Betlejewski P, Racine N, Ostrzycki A, Nawarawong W, Das S, Rouleau JL, Sopko G, Lee KL, Velazquez EJ, Panza JA. The association between blood pressure and long-term outcomes of patients with ischaemic cardiomyopathy with and without surgical revascularization: an analysis of the STICH trial. Eur Heart J. 2018 Oct 1;39(37):3464-3471. doi: 10.1093/eurheartj/ehy438. PMID 30113633
- [Derived] Stewart RAH, Szalewska D, Stebbins A, Al-Khalidi HR, Cleland JGH, Rynkiewicz A, Drazner MH, White HD, Mark DB, Roy A, Kosevic D, Rajda M, Jasinski M, Leng CY, Tungsubutra W, Desvigne-Nickens P, Velazquez EJ, Petrie MC. Six-minute walk distance after coronary artery bypass grafting compared with medical therapy in ischaemic cardiomyopathy. Open Heart. 2018 Feb 20;5(1):e000752. doi: 10.1136/openhrt-2017-000752. eCollection 2018. PMID 29531766
- [Derived] Pina IL, Zheng Q, She L, Szwed H, Lang IM, Farsky PS, Castelvecchio S, Biernat J, Paraforos A, Kosevic D, Favaloro LE, Nicolau JC, Varadarajan P, Velazquez EJ, Pai RG, Cyrille N, Lee KL, Desvigne-Nickens P; STICH Trial Investigators. Sex Difference in Patients With Ischemic Heart Failure Undergoing Surgical Revascularization: Results From the STICH Trial (Surgical Treatment for Ischemic Heart Failure). Circulation. 2018 Feb 20;137(8):771-780. doi: 10.1161/CIRCULATIONAHA.117.030526. PMID 29459462
- [Derived] Prior DL, Stevens SR, Holly TA, Krejca M, Paraforos A, Pohost GM, Byrd K, Kukulski T, Jones RH, Desvigne-Nickens P, Varadarajan P, Amanullah A, Lin G, Al-Khalidi HR, Aldea G, Santambrogio C, Bochenek A, Berman DS; STICH Trial Investigators. Regional left ventricular function does not predict survival in ischaemic cardiomyopathy after cardiac surgery. Heart. 2017 Sep;103(17):1359-1367. doi: 10.1136/heartjnl-2016-310693. Epub 2017 Apr 26. PMID 28446548
- [Derived] Petrie MC, Jhund PS, She L, Adlbrecht C, Doenst T, Panza JA, Hill JA, Lee KL, Rouleau JL, Prior DL, Ali IS, Maddury J, Golba KS, White HD, Carson P, Chrzanowski L, Romanov A, Miller AB, Velazquez EJ; STICH Trial Investigators. Ten-Year Outcomes After Coronary Artery Bypass Grafting According to Age in Patients With Heart Failure and Left Ventricular Systolic Dysfunction: An Analysis of the Extended Follow-Up of the STICH Trial (Surgical Treatment for Ischemic Heart Failure). Circulation. 2016 Nov 1;134(18):1314-1324. doi: 10.1161/CIRCULATIONAHA.116.024800. Epub 2016 Aug 29. PMID 27573034
- [Derived] Velazquez EJ, Lee KL, Jones RH, Al-Khalidi HR, Hill JA, Panza JA, Michler RE, Bonow RO, Doenst T, Petrie MC, Oh JK, She L, Moore VL, Desvigne-Nickens P, Sopko G, Rouleau JL; STICHES Investigators. Coronary-Artery Bypass Surgery in Patients with Ischemic Cardiomyopathy. N Engl J Med. 2016 Apr 21;374(16):1511-20. doi: 10.1056/NEJMoa1602001. Epub 2016 Apr 3. PMID 27040723
- [Derived] Jolicoeur EM, Dunning A, Castelvecchio S, Dabrowski R, Waclawiw MA, Petrie MC, Stewart R, Jhund PS, Desvigne-Nickens P, Panza JA, Bonow RO, Sun B, San TR, Al-Khalidi HR, Rouleau JL, Velazquez EJ, Cleland JGF. Importance of angina in patients with coronary disease, heart failure, and left ventricular systolic dysfunction: insights from STICH. J Am Coll Cardiol. 2015 Nov 10;66(19):2092-2100. doi: 10.1016/j.jacc.2015.08.882. PMID 26541919
- [Derived] Bonow RO, Castelvecchio S, Panza JA, Berman DS, Velazquez EJ, Michler RE, She L, Holly TA, Desvigne-Nickens P, Kosevic D, Rajda M, Chrzanowski L, Deja M, Lee KL, White H, Oh JK, Doenst T, Hill JA, Rouleau JL, Menicanti L; STICH Trial Investigators. Severity of Remodeling, Myocardial Viability, and Survival in Ischemic LV Dysfunction After Surgical Revascularization. JACC Cardiovasc Imaging. 2015 Oct;8(10):1121-1129. doi: 10.1016/j.jcmg.2015.03.013. Epub 2015 Sep 9. PMID 26363840
- [Derived] Wrobel K, Stevens SR, Jones RH, Selzman CH, Lamy A, Beaver TM, Djokovic LT, Wang N, Velazquez EJ, Sopko G, Kron IL, DiMaio JM, Michler RE, Lee KL, Yii M, Leng CY, Zembala M, Rouleau JL, Daly RC, Al-Khalidi HR. Influence of Baseline Characteristics, Operative Conduct, and Postoperative Course on 30-Day Outcomes of Coronary Artery Bypass Grafting Among Patients With Left Ventricular Dysfunction: Results From the Surgical Treatment for Ischemic Heart Failure (STICH) Trial. Circulation. 2015 Aug 25;132(8):720-30. doi: 10.1161/CIRCULATIONAHA.114.014932. PMID 26304663
- [Derived] MacDonald MR, She L, Doenst T, Binkley PF, Rouleau JL, Tan RS, Lee KL, Miller AB, Sopko G, Szalewska D, Waclawiw MA, Dabrowski R, Castelvecchio S, Adlbrecht C, Michler RE, Oh JK, Velazquez EJ, Petrie MC. Clinical characteristics and outcomes of patients with and without diabetes in the Surgical Treatment for Ischemic Heart Failure (STICH) trial. Eur J Heart Fail. 2015 Jul;17(7):725-34. doi: 10.1002/ejhf.288. Epub 2015 May 26. PMID 26011509
- [Derived] Mark DB, Knight JD, Velazquez EJ, Wasilewski J, Howlett JG, Smith PK, Spertus JA, Rajda M, Yadav R, Hamman BL, Malinowski M, Naik A, Rankin G, Harding TM, Drew LA, Desvigne-Nickens P, Anstrom KJ. Quality-of-life outcomes with coronary artery bypass graft surgery in ischemic left ventricular dysfunction: a randomized trial. Ann Intern Med. 2014 Sep 16;161(6):392-9. doi: 10.7326/M13-1380. PMID 25222386
- [Derived] Panza JA, Velazquez EJ, She L, Smith PK, Nicolau JC, Favaloro RR, Gradinac S, Chrzanowski L, Prabhakaran D, Howlett JG, Jasinski M, Hill JA, Szwed H, Larbalestier R, Desvigne-Nickens P, Jones RH, Lee KL, Rouleau JL. Extent of coronary and myocardial disease and benefit from surgical revascularization in ischemic LV dysfunction [Corrected]. J Am Coll Cardiol. 2014 Aug 12;64(6):553-61. doi: 10.1016/j.jacc.2014.04.064. PMID 25104523
- [Derived] Stewart RA, Szalewska D, She L, Lee KL, Drazner MH, Lubiszewska B, Kosevic D, Ruengsakulrach P, Nicolau JC, Coutu B, Choudhary SK, Mark DB, Cleland JG, Pina IL, Velazquez EJ, Rynkiewicz A, White H. Exercise capacity and mortality in patients with ischemic left ventricular dysfunction randomized to coronary artery bypass graft surgery or medical therapy: an analysis from the STICH trial (Surgical Treatment for Ischemic Heart Failure). JACC Heart Fail. 2014 Aug;2(4):335-43. doi: 10.1016/j.jchf.2014.02.009. Epub 2014 Jul 9. PMID 25023813
- [Derived] Doenst T, Cleland JG, Rouleau JL, She L, Wos S, Ohman EM, Krzeminska-Pakula M, Airan B, Jones RH, Siepe M, Sopko G, Velazquez EJ, Racine N, Gullestad L, Filgueira JL, Lee KL; STICH Investigators. Influence of crossover on mortality in a randomized study of revascularization in patients with systolic heart failure and coronary artery disease. Circ Heart Fail. 2013 May;6(3):443-50. doi: 10.1161/CIRCHEARTFAILURE.112.000130. Epub 2013 Mar 20. PMID 23515275
- [Derived] Panza JA, Holly TA, Asch FM, She L, Pellikka PA, Velazquez EJ, Lee KL, Borges-Neto S, Farsky PS, Jones RH, Berman DS, Bonow RO. Inducible myocardial ischemia and outcomes in patients with coronary artery disease and left ventricular dysfunction. J Am Coll Cardiol. 2013 May 7;61(18):1860-70. doi: 10.1016/j.jacc.2013.02.014. Epub 2013 Mar 7. PMID 23500234
- [Derived] Oh JK, Velazquez EJ, Menicanti L, Pohost GM, Bonow RO, Lin G, Hellkamp AS, Ferrazzi P, Wos S, Rao V, Berman D, Bochenek A, Cherniavsky A, Rogowski J, Rouleau JL, Lee KL; STICH Investigators. Influence of baseline left ventricular function on the clinical outcome of surgical ventricular reconstruction in patients with ischaemic cardiomyopathy. Eur Heart J. 2013 Jan;34(1):39-47. doi: 10.1093/eurheartj/ehs021. Epub 2012 May 14. PMID 22584648
- [Derived] Deja MA, Grayburn PA, Sun B, Rao V, She L, Krejca M, Jain AR, Leng Chua Y, Daly R, Senni M, Mokrzycki K, Menicanti L, Oh JK, Michler R, Wrobel K, Lamy A, Velazquez EJ, Lee KL, Jones RH. Influence of mitral regurgitation repair on survival in the surgical treatment for ischemic heart failure trial. Circulation. 2012 May 29;125(21):2639-48. doi: 10.1161/CIRCULATIONAHA.111.072256. Epub 2012 May 2. PMID 22553307
- [Derived] Bonow RO, Maurer G, Lee KL, Holly TA, Binkley PF, Desvigne-Nickens P, Drozdz J, Farsky PS, Feldman AM, Doenst T, Michler RE, Berman DS, Nicolau JC, Pellikka PA, Wrobel K, Alotti N, Asch FM, Favaloro LE, She L, Velazquez EJ, Jones RH, Panza JA; STICH Trial Investigators. Myocardial viability and survival in ischemic left ventricular dysfunction. N Engl J Med. 2011 Apr 28;364(17):1617-25. doi: 10.1056/NEJMoa1100358. Epub 2011 Apr 4. PMID 21463153
- [Derived] Velazquez EJ, Lee KL, Deja MA, Jain A, Sopko G, Marchenko A, Ali IS, Pohost G, Gradinac S, Abraham WT, Yii M, Prabhakaran D, Szwed H, Ferrazzi P, Petrie MC, O'Connor CM, Panchavinnin P, She L, Bonow RO, Rankin GR, Jones RH, Rouleau JL; STICH Investigators. Coronary-artery bypass surgery in patients with left ventricular dysfunction. N Engl J Med. 2011 Apr 28;364(17):1607-16. doi: 10.1056/NEJMoa1100356. Epub 2011 Apr 4. PMID 21463150
- [Derived] Zembala M, Michler RE, Rynkiewicz A, Huynh T, She L, Lubiszewska B, Hill JA, Jandova R, Dagenais F, Peterson ED, Jones RH. Clinical characteristics of patients undergoing surgical ventricular reconstruction by choice and by randomization. J Am Coll Cardiol. 2010 Aug 3;56(6):499-507. doi: 10.1016/j.jacc.2010.03.054. PMID 20670761
- [Derived] Jones RH, White H, Velazquez EJ, Shaw LK, Pietrobon R, Panza JA, Bonow RO, Sopko G, O'Connor CM, Rouleau JL. STICH (Surgical Treatment for Ischemic Heart Failure) trial enrollment. J Am Coll Cardiol. 2010 Aug 3;56(6):490-8. doi: 10.1016/j.jacc.2009.11.102. PMID 20670760
- [Derived] Mark DB, Knight JD, Velazquez EJ, Howlett JG, Spertus JA, Djokovic LT, Harding TM, Rankin GR, Drew LA, Szygula-Jurkiewicz B, Adlbrecht C, Anstrom KJ; Surgical Treatment for Ischemic Heart Failure (STICH) Trial Investigators. Quality of life and economic outcomes with surgical ventricular reconstruction in ischemic heart failure: results from the Surgical Treatment for Ischemic Heart Failure trial. Am Heart J. 2009 May;157(5):837-44, 844.e1-3. doi: 10.1016/j.ahj.2009.03.008. Epub 2009 Apr 1. PMID 19376309
- [Derived] Jones RH, Velazquez EJ, Michler RE, Sopko G, Oh JK, O'Connor CM, Hill JA, Menicanti L, Sadowski Z, Desvigne-Nickens P, Rouleau JL, Lee KL; STICH Hypothesis 2 Investigators. Coronary bypass surgery with or without surgical ventricular reconstruction. N Engl J Med. 2009 Apr 23;360(17):1705-17. doi: 10.1056/NEJMoa0900559. Epub 2009 Mar 29. PMID 19329820
- See also: STICH trial website — http://www.stichtrial.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pts were assigned to 1 of 3 strata before randomization. All pts in stratum C and some pts in stratum B were randomly assigned to med therapy + CABG or med therapy + CABG + SVR (Hypothesis 2 component of the trial-HO2). 76 of stratum B pts who were randomized to med therapy + CABG group belong to both H01 and H02.
Pre-assignment Details: Stratum A: eligible for med. therapy alone or med therapy + CABG; Stratum C: eligible for med therapy + CABG or med therapy + CABG + SVR; Stratum B: eligible for all 3 treatment options. All pts in stratum A and some of the pts in stratum B were randomized to either med therapy alone or med therapy + CABG (Hypothesis 1 of the STICH trial--H01).
Groups:
- H01: Medication: 50% of H01 patients were randomized to this medical therapy alone arm. Throughout the trial follow-up period, the use of guideline-recommended medications and devices for the treatment of heart failure and CAD was strongly emphasized for all patients in this treatment arm.
- H01: Medication + CABG: 50% of H01 patients were randomized to medical therapy plus CABG arm. In addition to the guideline-recommended medications, coronary artery bypass graft (CABG) surgery was to be performed for patients randomized to this treatment arm. This group does not include those 76 patients who belong to both H01 and H02.
- H01+H02: Medication + CABG: This group includes those 76 patients who belong to both H01 and H02. These patients were randomized to medical therapy plus CABG arm. In addition to the guideline-recommended medications, coronary artery bypass graft (CABG) surgery was to be performed for patients randomized to this treatment arm.
- H02: Medication+CABG: 50% of H02 patients were randomized to this medical therapy plus CABG arm. In addition to the guideline-recommended medications, coronary artery bypass graft (CABG) surgery was to be performed for patients randomized to this treatment arm. This group does not include those 76 patients who belong to both H01 and H02.
- H02: Medication+CABG+SVR: 50% of H02 patients were randomized to this medical therapy plus CABG plus SVR arm. In addition to the guideline-recommended medications, both the coronary artery bypass graft (CABG) surgery and the surgical ventricular reconstruction (SVR) were to be performed for patients randomized to this treatment arm.
Period: 5 Year Follow up
Arm/Group | H01: Medication | H01: Medication + CABG | H01+H02: Medication + CABG | H02: Medication+CABG | H02: Medication+CABG+SVR
Started | 602 | 534 | 76 | 423 (76 of stratum B pts who were randomized to med therapy + CABG group belong to both H01 and H02.) | 501
Completed | 600 | 532 | 75 | 416 | 498
Not Completed | 2 | 2 | 1 | 7 | 3
Not completed — Lost to Follow-up | 2 | 2 | 1 | 7 | 3
Period: 10 Year Follow up
Arm/Group | H01: Medication | H01: Medication + CABG | H01+H02: Medication + CABG | H02: Medication+CABG | H02: Medication+CABG+SVR
Started | 602 (all participants who started H01 were counted as starting the 10 year follow up.) | 534 (all participants who started H01 were counted as starting the 10 year follow up.) | 76 (all participants who started H01 were counted as starting the 10 year follow up.) | 0 (H02 arm was not extended and ended at year 5) | 0 (H02 arm was not extended and ended at year 5)
Completed | 590 | 524 | 73 | 0 (H02 arm was not extended and ended at year 5) | 0 (H02 arm was not extended and ended at year 5)
Not Completed | 12 | 10 | 3 | 0 | 0
Not completed — Lost to Follow-up | 12 | 10 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H01: Medication | H01: Medication + CABG | H01+H02: Medication + CABG | H02: Medication+CABG | H02: Medication+CABG+SVR | Total
Number analyzed (Participants) | 602 | 534 | 76 | 423 | 501 | 2136
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [53 to 67] | 60 [54 to 68] | 61 [54 to 68] | 62 [55 to 69] | 62 [55 to 69] | 60 [54 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 64 | 9 | 69 | 69 | 286
  Male | 527 | 470 | 67 | 354 | 432 | 1850

OUTCOME MEASURES:

1. Primary Outcome: H01: All Cause Mortality
Time Frame: 5 years post randomization
Population: The Total H01: Medication + CABG group includes the H01: Medication + CABG group and those 76 patients who belong to H01+H02: Medication + CABG arm.
Measure: Number; unit: participants
Groups:
- H01: Medication: H01 patients were randomized to medical therapy alone. Throughout the trial follow-up period, the use of guideline-recommended medications and devices for the treatment of heart failure and CAD was strongly emphasized for all patients in this treatment arm.
- Total H01: Medication + CABG: H01 patients were randomized to medical therapy plus CABG. In addition to the guideline-recommended medications, coronary artery bypass graft (CABG) surgery was to be performed for patients randomized to this treatment arm.
  The Total H01: Medication + CABG group includes the H01: Medication + CABG group and those 76 patients who belong to H01+H02: Medication + CABG arm.
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 244 | 218
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p = 0.12, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.72 to 1.04] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

2. Primary Outcome: H01: All Cause Mortality
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 398 | 359
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p = 0.02, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.73 to 0.97] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

3. Primary Outcome: H02: All-cause Mortality or Cardiovascular Hospitalization
Time Frame: 5 years post randomization
Population: The Total H02: Medication + CABG group includes the H02: Medication + CABG group and those 76 patients who belong to H01+H02: Medication + CABG arm.
Measure: Number; unit: participants
Groups:
- Total H02: Medication+CABG: H02 patients were randomized to medical therapy plus CABG arm. In addition to the guideline-recommended medications, coronary artery bypass graft (CABG) surgery was to be performed for patients randomized to this treatment arm.
  The Total H02: Medication + CABG group includes the H02: Medication + CABG group and those 76 patients who belong to H01+H02: Medication + CABG arm.
Arm/Group | H02: Medication+CABG+SVR | Total H02: Medication+CABG
Number analyzed (Participants) | 501 | 499
participants | 289 | 292
Statistical Analysis 1: Comparison: H02: Medication+CABG+SVR vs Total H02: Medication+CABG; Test type: Superiority or Other; p = 0.90, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.84 to 1.17] — Hazard Ratio is for (H02: Medication + CABG + SVR) versus (H02: Medication + CABG)

4. Secondary Outcome: H01: Cardiovascular Mortality (Defined as Sudden Death or Death Attributed to Recurrent MI, HF, a Cardiovascular Procedure, Stroke, or Other Cardiovascular Etiology).
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 610 | 602
participants | 247 | 297
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority or Other; p = 0.006, Log Rank; Hazard Ratio, log = 0.79, 95% CI 2-sided [0.66 to 0.93] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

5. Secondary Outcome: H01: Cardiovascular Mortality (Defined as Sudden Death or Death Attributed to Recurrent MI, HF, a Cardiovascular Procedure, Stroke, or Other Cardiovascular Etiology).
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 610 | 602
participants | 168 | 201
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority or Other; p = 0.05, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.66 to 1.00] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

6. Secondary Outcome: H01: Mortality or Cardiovascular Hospitalization
Time Frame: up to 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 411 | 351
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.64 to 0.85] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

7. Secondary Outcome: H01: Mortality or Cardiovascular Hospitalization
Time Frame: up to 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 524 | 467
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.64 to 0.82] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

8. Secondary Outcome: H02: All-cause Mortality
Time Frame: up to 5 years
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 141 | 138
Statistical Analysis 1: Comparison: Total H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority or Other; p = 0.98, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.79 to 1.26] — Hazard Ratio is for (H02: Medication + CABG + SVR) versus (H02: Medication + CABG)

9. Secondary Outcome: H01: All-cause Mortality Within 30 Days After Randomization
Time Frame: 30 days post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 7 | 22
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.35 to 7.52] — Odds Ratio is for (H01: Medication +CABG) versus (H01: Medication)

10. Secondary Outcome: H02: All-cause Mortality Within 30 Days After Randomization
Time Frame: 30 days post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 22 | 30
Statistical Analysis 1: Comparison: Total H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority or Other; p = 0.275, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.78 to 2.41] — Odds Ratio is for (H02: Medication + CABG + SVR) versus (H02: Medication + CABG)

11. Secondary Outcome: H01: All-cause Mortality or Heart-failure Hospitalization
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 324 | 290
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p = 0.030, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 0.98] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

12. Secondary Outcome: H02: All-cause Mortality or Heart-failure Hospitalization
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 211 | 214
Statistical Analysis 1: Comparison: Total H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority or Other; p = 0.401, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.89 to 1.31] — Hazard Ratio is for (H02: Medication + CABG + SVR) versus (H02: Medication + CABG)

13. Secondary Outcome: H01: All-cause Mortality or Heart-failure Hospitalization
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 450 | 404
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p = 0.002, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.71 to 0.93] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

14. Secondary Outcome: H01: Heart Failure Hospitalization
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 169 | 127

15. Secondary Outcome: H02: Heart Failure Hospitalization
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 95 | 99

16. Secondary Outcome: H01: Heart Failure Hospitalization
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 201 | 157

17. Secondary Outcome: H01: Cardiac Procedure: Heart Transplant
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 3 | 0

18. Secondary Outcome: H02: Cardiac Procedure: Heart Transplant
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 2 | 7

19. Secondary Outcome: H01: Cardiac Procedure: Heart Transplant
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 4 | 1

20. Secondary Outcome: H01: Cardiac Procedure: Left Ventricular Assist Device (LVAD)
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 2 | 2

21. Secondary Outcome: H02: Cardiac Procedure: Left Ventricular Assist Device (LVAD)
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 2 | 2

22. Secondary Outcome: H01: Cardiac Procedure: Left Ventricular Assist Device (LVAD)
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 2 | 4

23. Secondary Outcome: H01: Cardiac Procedure: Implantable Cardioverter Defibrillator (ICD)
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 98 | 76

24. Secondary Outcome: H02: Cardiac Procedure: Implantable Cardioverter Defibrillator (ICD)
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 100 | 86

25. Secondary Outcome: H01: Cardiac Procedure: Implantable Cardioverter Defibrillator (ICD)
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 118 | 105

26. Secondary Outcome: H01: Stroke
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 34 | 41

27. Secondary Outcome: H01: Stroke
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 41 | 47

28. Secondary Outcome: H02: Stroke
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 31 | 23

29. Secondary Outcome: H01: All-cause Mortality or Revascularization (CABG or PCI)
Description: CABG = coronary artery bypass grafting. For patients randomized to CABG or CABG +SVR group, this represents the repeat CABG received during follow-up. PCI = Percutaneous Coronary Intervention.
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 333 | 237
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.51 to 0.71] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

30. Secondary Outcome: H02: All-cause Mortality or Revascularization (CABG or PCI)
Description: as for outcome 29
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 174 | 152
Statistical Analysis 1: Comparison: Total H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority or Other; p = 0.414, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.73 to 1.13] — Hazard Ratio is for (H02: Medication + CABG + SVR) versus (H02: Medication + CABG)

31. Secondary Outcome: H01: All-cause Mortality or Revascularization (CABG or PCI)
Description: as for outcome 29
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 478 | 388
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.55 to 0.73] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

32. Secondary Outcome: H01: All-cause Mortality, Heart Transplant or LVAD
Description: LVAD=Left Ventricular Assist Device
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 245 | 218
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p = 0.108, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.72 to 1.03] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

33. Secondary Outcome: H02: All-cause Mortality, Heart Transplant or LVAD
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 148 | 145
Statistical Analysis 1: Comparison: Total H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority or Other; p = 0.717, Log Rank; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.83 to 1.32] — Hazard Ratio is for (H02: Medication + CABG + SVR) versus (H02: Medication + CABG)

34. Secondary Outcome: H01: All-cause Mortality, Heart Transplant or LVAD
Description: LVAD=Left Ventricular Assist Device
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 400 | 361
Statistical Analysis 1: Comparison: H01: Medication vs Total H01: Medication + CABG; Test type: Superiority or Other; p = 0.018, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.73 to 0.97] — Hazard Ratio is for (H01: Medication +CABG) versus (H01: Medication)

35. Secondary Outcome: H01: All-cause (Unplanned and Elective) Hospitalization
Time Frame: 5 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 340 | 290

36. Secondary Outcome: H02: All-cause (Unplanned and Elective) Hospitalization
Time Frame: 5 years post randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 499 | 501
participants | 272 | 268

37. Secondary Outcome: H01: All-cause (Unplanned and Elective) Hospitalization
Time Frame: 10 years post randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 602 | 610
participants | 383 | 349

38. Secondary Outcome: H01: 6 Minute Walk Distance
Time Frame: From randomization to 24 month follow-up
Population: Only patients with 6-minute walk distance data at baseline, 4 months or 24 months were analyzed.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 559 | 552
meters
  Baseline: number analyzed (Participants) | 535 | 506
  Baseline | 333.97 (117.76) | 333.04 (117.06)
  4 month: number analyzed (Participants) | 442 | 404
  4 month | 364.25 (111.24) | 376.46 (118.87)
  Changed from baseline to 4 months: number analyzed (Participants) | 420 | 368
  Changed from baseline to 4 months | 28.2 (102.44) | 37.76 (108.93)
  24 month: number analyzed (Participants) | 301 | 296
  24 month | 381.55 (120.86) | 377.84 (122.62)
  Change from baseline to 24 Months: number analyzed (Participants) | 287 | 264
  Change from baseline to 24 Months | 34.11 (112.9) | 31.18 (128.99)

39. Secondary Outcome: H02: 6 Minute Walk Distance
Time Frame: From randomization to 24 month follow-up
Population: Only patients with 6-minute walk distance data at baseline, 4 months or 24 months were analyzed.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 420 | 429
meters
  Baseline: number analyzed (Participants) | 335 | 357
  Baseline | 339.38 (126.11) | 357.23 (116.91)
  4 month: number analyzed (Participants) | 335 | 341
  4 month | 385.89 (123.49) | 407.03 (121.38)
  Changed from baseline to 4 months: number analyzed (Participants) | 259 | 273
  Changed from baseline to 4 months | 44.42 (122.64) | 46.09 (113.67)
  24 month: number analyzed (Participants) | 256 | 248
  24 month | 400.66 (121.67) | 425.18 (121.46)
  Change from baseline to 24 Months: number analyzed (Participants) | 196 | 206
  Change from baseline to 24 Months | 51.51 (125.65) | 55.6 (112.66)

40. Secondary Outcome: H01: Exercise Duration
Description: Record the total duration of exercise in minutes and seconds for patients performing the modified Bruce exercise treadmill test
Time Frame: From randomization to 24 months follow-up
Population: Only patients with exercise duration data at baseline or 24 months were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 269 | 242
minutes
  Baseline: number analyzed (Participants) | 256 | 230
  Baseline | 6.85 (3.4) | 6.3 (3.39)
  24 month: number analyzed (Participants) | 118 | 117
  24 month | 7.78 (3.32) | 7.97 (3.32)
  Change from baseline to 24 Months: number analyzed (Participants) | 105 | 105
  Change from baseline to 24 Months | 0.71 (3.51) | 0.83 (3.26)

41. Secondary Outcome: H02: Exercise Duration
Description: as for outcome 40
Time Frame: From randomization to 24 months follow-up
Population: Only patients with exercise duration data at baseline or 24 months were analyzed.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 119 | 138
meters
  Baseline: number analyzed (Participants) | 106 | 127
  Baseline | 6.19 (3.42) | 7.16 (3.47)
  24 month: number analyzed (Participants) | 62 | 67
  24 month | 7.67 (3.3) | 8.41 (3.41)
  Change from baseline to 24 Months: number analyzed (Participants) | 49 | 56
  Change from baseline to 24 Months | 1.15 (3.01) | 0.47 (3.42)

42. Secondary Outcome: H01: LVEF by ECHO Core Lab During Follow-up
Description: Left ventricular ejection fraction (LVEF) measured by Echocardiography (ECHO) core lab
Time Frame: From randomization to 24 months follow-up
Population: Only patients with ECHO LVEF data at baseline, 4 months or 24 months were analyzed.
Measure: Mean (Standard Deviation); unit: Percent ejection fraction
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 584 | 589
Percent ejection fraction
  Baseline: number analyzed (Participants) | 566 | 558
  Baseline | 28.69 (8.33) | 28.43 (8.24)
  4 month: number analyzed (Participants) | 461 | 436
  4 month | 30.83 (9.41) | 30.66 (10.73)
  Changed from baseline to 4 months: number analyzed (Participants) | 447 | 410
  Changed from baseline to 4 months | 2.21 (8.8) | 2.06 (10.06)
  24 month: number analyzed (Participants) | 327 | 320
  24 month | 31.39 (10.75) | 31.15 (11.14)
  Change from baseline to 24 Months: number analyzed (Participants) | 319 | 301
  Change from baseline to 24 Months | 2.2 (11.31) | 2.22 (10.67)

43. Secondary Outcome: H02: LVEF by ECHO Core Lab During Follow-up
Description: Left ventricular ejection fraction (LVEF) measured by Echocardiography (ECHO) core lab
Time Frame: From randomization to 24 months follow-up
Population: Only patients with ECHO LVEF data at baseline, 4 months or 24 months were analyzed.
Measure: Mean (Standard Deviation); unit: Percent ejection fraction
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 484 | 484
Percent ejection fraction
  Baseline: number analyzed (Participants) | 464 | 464
  Baseline | 29.13 (7.74) | 29.49 (8.23)
  4 month: number analyzed (Participants) | 378 | 359
  4 month | 31.47 (10.4) | 33.35 (9.79)
  Changed from baseline to 4 months: number analyzed (Participants) | 361 | 341
  Changed from baseline to 4 months | 2.16 (10.23) | 3.04 (9.7)
  24 month: number analyzed (Participants) | 289 | 275
  24 month | 31.89 (11.38) | 33.55 (10.91)
  Change from baseline to 24 Months: number analyzed (Participants) | 277 | 264
  Change from baseline to 24 Months | 2.24 (11.11) | 2.93 (10.95)

44. Secondary Outcome: H01: LVEF by RN Core Lab During Follow-up
Description: Left ventricular ejection fraction (LVEF) measured by radionuclide (RN) core lab.
Time Frame: From randomization to 24 months follow-up
Population: Only patients with RN LVEF data at Baseline, 4-months or 24-months were analyzed.
Measure: Mean (Standard Deviation); unit: Percent ejection fraction
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 250 | 255
Percent ejection fraction
  Baseline: number analyzed (Participants) | 241 | 242
  Baseline | 26.83 (8.66) | 26.66 (8.41)
  4 month: number analyzed (Participants) | 56 | 55
  4 month | 27.2 (9.5) | 27.81 (9.73)
  Changed from baseline to 4 months: number analyzed (Participants) | 50 | 44
  Changed from baseline to 4 months | 0.99 (5.88) | 2.65 (6.36)
  24 month: number analyzed (Participants) | 26 | 28
  24 month | 30.65 (10.74) | 27.79 (9.05)
  Change from baseline to 24 Months: number analyzed (Participants) | 21 | 23
  Change from baseline to 24 Months | 3.99 (8.24) | 1.77 (5.63)

45. Secondary Outcome: H02: LVEF by RN Core Lab During Follow-up
Description: Left ventricular ejection fraction (LVEF) measured by radionuclide (RN) core lab.
Time Frame: From randomization to 24 months follow-up
Population: Only patients with RN LVEF data at Baseline, 4-months or 24-months were analyzed.
Measure: Mean (Standard Deviation); unit: Percent ejection fraction
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 214 | 216
Percent ejection fraction
  Baseline: number analyzed (Participants) | 168 | 182
  Baseline | 27.14 (8.18) | 26.55 (7.83)
  4 month: number analyzed (Participants) | 132 | 148
  4 month | 30.65 (10.41) | 33.5 (9.42)
  Changed from baseline to 4 months: number analyzed (Participants) | 98 | 123
  Changed from baseline to 4 months | 2.23 (7.11) | 6.49 (7.91)
  24 month: number analyzed (Participants) | 95 | 95
  24 month | 29.95 (10.97) | 34.2 (10.3)
  Change from baseline to 24 Months: number analyzed (Participants) | 69 | 78
  Change from baseline to 24 Months | 2.01 (9.58) | 6.79 (9.12)

46. Secondary Outcome: H01: LVEF by CMR Core Lab During Follow-up
Description: Left ventricular ejection fraction (LVEF) measured by cardiovascular magnetic resonance (CMR) core lab.
Time Frame: From randomization to 24 months follow-up
Population: Only patients with CMR LVEF data at baseline, 4 months or 24 months were analyzed.
Measure: Mean (Standard Deviation); unit: Percent ejection fraction
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 50 | 68
Percent ejection fraction
  Baseline: number analyzed (Participants) | 46 | 64
  Baseline | 29.51 (11.02) | 23.35 (9.49)
  4 month: number analyzed (Participants) | 25 | 27
  4 month | 28.6 (11.11) | 28.63 (13.16)
  Changed from baseline to 4 months: number analyzed (Participants) | 21 | 24
  Changed from baseline to 4 months | 0.07 (8.82) | 2.85 (12.87)
  24 month: number analyzed (Participants) | 11 | 12
  24 month | 32.72 (14.7) | 31.47 (9.06)
  Change from baseline to 24 Months: number analyzed (Participants) | 10 | 10
  Change from baseline to 24 Months | -1.09 (10.63) | 2.13 (13.27)

47. Secondary Outcome: H02: LVEF by CMR Core Lab During Follow-up
Description: Left ventricular ejection fraction (LVEF) measured by cardiovascular magnetic resonance (CMR) core lab.
Time Frame: From randomization to 24 months follow-up
Population: Only patients with CMR LVEF data at baseline, 4 months or 24 months were analyzed.
Measure: Mean (Standard Deviation); unit: Percent ejection fraction
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 207 | 196
Percent ejection fraction
  Baseline: number analyzed (Participants) | 184 | 171
  Baseline | 27.82 (10.26) | 27.25 (11.47)
  4 month: number analyzed (Participants) | 120 | 115
  4 month | 31.65 (13.53) | 34.37 (13.41)
  Changed from baseline to 4 months: number analyzed (Participants) | 101 | 97
  Changed from baseline to 4 months | 2.84 (11.86) | 7.1 (11.86)
  24 month: number analyzed (Participants) | 50 | 60
  24 month | 28.46 (10.57) | 33.1 (13.79)
  Change from baseline to 24 Months: number analyzed (Participants) | 40 | 48
  Change from baseline to 24 Months | -0.51 (14.61) | 5.39 (13.23)

48. Secondary Outcome: H01: B-type Natriuretic Peptide (BNP)
Description: B-type natriuretic peptide (BNP) by Neurohormonal/cytokine/genetic (NCG) core lab during follow-up
Time Frame: From randomization to 24 months follow-up
Population: Only patients with BNP data at baseline or 4 months were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | H01: Medication | Total H01: Medication + CABG
Number analyzed (Participants) | 314 | 325
pg/mL
  Baseline: number analyzed (Participants) | 297 | 310
  Baseline | 497.29 (627.49) | 478.73 (521.11)
  4 month: number analyzed (Participants) | 259 | 249
  4 month | 408.69 (413.27) | 484.39 (554.42)
  Changed from baseline to 4 months: number analyzed (Participants) | 242 | 234
  Changed from baseline to 4 months | -20.65 (405.44) | 33.37 (566.62)

49. Secondary Outcome: H02: B-type Natriuretic Peptide (BNP)
Description: B-type natriuretic peptide (BNP) by Neurohormonal/cytokine/genetic (NCG) core lab during follow-up
Time Frame: From randomization to 24 months follow-up
Population: Only patients with BNP data at baseline or 4 months were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Total H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 386 | 392
pg/mL
  Baseline | 453.73 (563.1) | 452.45 (665.06)
  4 month: number analyzed (Participants) | 296 | 306
  4 month | 460.14 (508.35) | 467.83 (579.42)
  Changed from baseline to 4 months: number analyzed (Participants) | 276 | 285
  Changed from baseline to 4 months | 19.75 (600.26) | 72.23 (554.2)

50. Secondary Outcome: H01: SF-36 Mental Health Subscale
Description: Short Form 36 Health Status Questionnaire (SF-36) Mental Health Subscale: These 5 items assess anxiety, depression, emotional control, and psychological well-being. Response choices range from "All of the time" (1) to "None of the time" (6). Item values are summed and then transformed to a 0-100 scale where higher scores indicate better mental health. (Final scores are normalized to a mean of 50 and standard deviation of 10.)
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 597 | 584
units on a scale
  Baseline | 43.7 (11.8) | 44.4 (11.8)
  4 Months: number analyzed (Participants) | 503 | 521
  4 Months | 48.2 (10.2) | 47.2 (11.2)
  12 Months: number analyzed (Participants) | 456 | 454
  12 Months | 48.8 (11.1) | 47.0 (11.8)
  24 Months: number analyzed (Participants) | 398 | 403
  24 Months | 48.6 (10.5) | 46.8 (11.8)
  36 Months: number analyzed (Participants) | 392 | 372
  36 Months | 48.5 (11.1) | 48.2 (10.8)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.015, Chi-squared — 4 months; H01 P-values were based on the Chi-Square test applied to maximum likelihood estimates derived from an adjusted mixed model
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.002, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.011, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.44, Chi-squared — 36 months

51. Secondary Outcome: H02: SF-36 Mental Health Subscale
Description: These 5 items assess anxiety, depression, emotional control, and psychological well-being. Response choices range from "All of the time" (1) to "None of the time" (6). Item values are summed and then transformed to a 0-100 scale where higher scores indicate better mental health. (Final scores are normalized to a mean of 50 and standard deviation of 10.)
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 489 | 481
units on a scale
  Baseline | 41 [32 to 50] | 41 [35 to 50]
  4 Months: number analyzed (Participants) | 410 | 407
  4 Months | 50 [39 to 57] | 50 [41 to 57]
  12 Months: number analyzed (Participants) | 380 | 389
  12 Months | 53 [44 to 60] | 50 [41 to 57]
  24 Months: number analyzed (Participants) | 345 | 347
  24 Months | 50 [41 to 57] | 50 [41 to 57]
  36 Months: number analyzed (Participants) | 310 | 313
  36 Months | 50 [41 to 60] | 50 [44 to 57]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)

52. Secondary Outcome: H01:SF-36 Role Physical Subscale
Description: These 4 items assess limitations and difficulty performing work or other usual activities as a result of one's physical health. Response choices are either "Yes" (1) or "No" (2). Item values are summed and then transformed to a 0-100 scale where higher scores indicate better outcomes. (Final scores are normalized to a mean of 50 and standard deviation of 10.)
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 581 | 569
units on a scale
  Baseline | 36.1 (10.9) | 36.6 (11.2)
  4 Months: number analyzed (Participants) | 486 | 508
  4 Months | 43.0 (11.8) | 42.6 (11.8)
  12 Months: number analyzed (Participants) | 445 | 446
  12 Months | 45.7 (11.4) | 43.1 (12.2)
  24 Months: number analyzed (Participants) | 396 | 394
  24 Months | 46.6 (11.4) | 44.7 (12.2)
  36 Months: number analyzed (Participants) | 388 | 368
  36 Months | 46.0 (11.2) | 44.8 (11.6)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.31, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.002, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority — 24 months; p = 0.028, Chi-squared
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.079, Chi-squared — 36 months

53. Secondary Outcome: H02: SF-36 Role Physical Subscale
Description: as for outcome 52
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 466 | 466
units on a scale
  Baseline | 28 [28 to 35] | 28 [28 to 42]
  4 Months: number analyzed (Participants) | 400 | 393
  4 Months | 42 [28 to 56] | 42 [28 to 56]
  12 Months: number analyzed (Participants) | 372 | 389
  12 Months | 49 [35 to 56] | 49 [35 to 56]
  24 Months: number analyzed (Participants) | 340 | 339
  24 Months | 49 [28 to 56] | 49 [35 to 56]
  36 Months: number analyzed (Participants) | 308 | 309
  36 Months | 49 [35 to 56] | 56 [35 to 56]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.61, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney) — 36 months

54. Secondary Outcome: H01:SF-36 Role Emotional Subscale
Description: These 3 items assess limitations and difficulty performing work or other usual activities as a result of any emotional problems (such as feeling depressed or anxious). Response choices are either "Yes" (1) or "No" (2). Item values are summed and then transformed to a 0-100 scale where higher scores indicate better outcomes. (Final scores are normalized to a mean of 50 and standard deviation of 10.)
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 588 | 582
units on a scale
  Baseline | 39.0 (14.2) | 40.0 (14.4)
  4 Months: number analyzed (Participants) | 499 | 511
  4 Months | 45.3 (13.2) | 44.6 (13.4)
  12 Months: number analyzed (Participants) | 455 | 450
  12 Months | 46.4 (12.8) | 45.9 (13.3)
  24 Months: number analyzed (Participants) | 398 | 396
  24 Months | 47.5 (12.1) | 46.8 (12.8)
  36 Months: number analyzed (Participants) | 392 | 364
  36 Months | 48.0 (11.8) | 47.0 (12.4)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.063, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.187, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.168, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.050, Chi-squared — 36 months

55. Secondary Outcome: H02: SF-36 Role Emotional Subscale
Description: as for outcome 54
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 482 | 477
units on a scale
  Baseline | 34 [24 to 55] | 34 [24 to 55]
  4 Months: number analyzed (Participants) | 409 | 402
  4 Months | 55 [34 to 55] | 55 [34 to 55]
  12 Months: number analyzed (Participants) | 377 | 384
  12 Months | 55 [45 to 55] | 55 [45 to 55]
  24 Months: number analyzed (Participants) | 341 | 344
  24 Months | 55 [45 to 55] | 55 [34 to 55]
  36 Months: number analyzed (Participants) | 306 | 308
  36 Months | 55 [45 to 55] | 55 [45 to 55]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney) — 36 months

56. Secondary Outcome: H01:SF-36 Social Functioning Subscale
Description: These 2 items assess the limitations on social activities with others. Response choices range from "Extremely" or "All of the time" (1) to "Not at all" or "None of the time" (5). Item values are summed and then transformed to a 0-100 scale where higher scores indicate better social functioning. (Final scores are normalized to a mean of 50 and standard deviation of 10.)
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 601 | 588
units on a scale
  Baseline | 41.8 (12.0) | 42.1 (12.0)
  4 Months: number analyzed (Participants) | 505 | 523
  4 Months | 47.0 (11.1) | 45.8 (11.3)
  12 Months: number analyzed (Participants) | 457 | 456
  12 Months | 48.7 (10.4) | 46.1 (11.7)
  24 Months: number analyzed (Participants) | 401 | 403
  24 Months | 48.3 (9.9) | 46.1 (11.1)
  36 Months: number analyzed (Participants) | 394 | 370
  36 Months | 47.8 (10.3) | 47.1 (10.2)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.039, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.002, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.008, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.31, Chi-squared — 36 months

57. Secondary Outcome: H02: SF-36 Social Functioning Subscale
Description: as for outcome 56
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 490 | 485
units on a scale
  Baseline | 41 [30 to 52] | 35 [30 to 46]
  4 Months: number analyzed (Participants) | 410 | 411
  4 Months | 52 [35 to 57] | 52 [41 to 57]
  12 Months: number analyzed (Participants) | 380 | 389
  12 Months | 52 [41 to 57] | 52 [41 to 57]
  24 Months: number analyzed (Participants) | 345 | 349
  24 Months | 52 [41 to 57] | 52 [41 to 57]
  36 Months: number analyzed (Participants) | 308 | 313
  36 Months | 52 [41 to 57] | 52 [41 to 57]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney) — 36 months

58. Secondary Outcome: H01:SF-36 Vitality Subscale
Description: These 4 items assess energy level and fatigue. Response choices range from "All of the time" (1) to "None of the time" (6). Item values are summed and then transformed to a 0-100 scale where higher scores indicate better vitality. (Final scores are normalized to a mean of 50 and standard deviation of 10.)
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 598 | 586
units on a scale
  Baseline | 46.4 (10.3) | 47.5 (10.9)
  4 Months: number analyzed (Participants) | 503 | 522
  4 Months | 51.6 (9.8) | 50.5 (10.5)
  12 Months: number analyzed (Participants) | 456 | 453
  12 Months | 52.2 (10.1) | 49.9 (10.9)
  24 Months: number analyzed (Participants) | 398 | 403
  24 Months | 51.9 (9.9) | 49.4 (10.5)
  36 Months: number analyzed (Participants) | 393 | 372
  36 Months | 51.4 (10.0) | 50.6 (10.4)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 4 months
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.024, Chi-squared — 36 months

59. Secondary Outcome: H02: SF-36 Vitality Subscale
Description: as for outcome 58
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 489 | 480
units on a scale
  Baseline | 44 [37 to 51] | 44 [37 to 49]
  4 Months: number analyzed (Participants) | 410 | 409
  4 Months | 51 [42 to 59] | 51 [44 to 59]
  12 Months: number analyzed (Participants) | 380 | 390
  12 Months | 53 [44 to 59] | 51 [44 to 59]
  24 Months: number analyzed (Participants) | 345 | 347
  24 Months | 51 [44 to 59] | 51 [44 to 61]
  36 Months: number analyzed (Participants) | 309 | 313
  36 Months | 51 [44 to 59] | 51 [44 to 61]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney) — 36 months

60. Secondary Outcome: H01:SF-12 Physical Component Summary (PCS) Scale
Description: Twelve items that reflect both physical and mental health are selected from the SF-36 subscales and combined according to an algebraic formula using published weights and constants: (a) First, the items are coded so that a higher value indicates better health; (b) then indicator variables (1/0) are created for the item response choice categories; (c) next, the 35 indicator variables are weighted using "physical" regression weights from the general US population and summed to produce the PCS-12 score; and (d) finally, a normalized score (with a mean of 50 and standard deviation of 10) is obtained by adding the "physical" constant from the scoring table to the sum of the 35 products.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 534 | 530
units on a scale
  Baseline | 37.8 (6.1) | 38.4 (5.7)
  4 Months: number analyzed (Participants) | 448 | 455
  4 Months | 40.2 (5.9) | 39.9 (5.8)
  12 Months: number analyzed (Participants) | 403 | 405
  12 Months | 41.0 (5.3) | 40.0 (6.0)
  24 Months: number analyzed (Participants) | 370 | 356
  24 Months | 41.3 (5.7) | 40.9 (5.8)
  36 Months: number analyzed (Participants) | 347 | 333
  36 Months | 40.8 (5.5) | 41.3 (5.8)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.051, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.003, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.065, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.83, Chi-squared — 36 months

61. Secondary Outcome: H02: SF-12 Physical Component Summary (PCS) Scale
Description: as for outcome 60
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 433 | 426
units on a scale
  Baseline | 37 [33 to 41] | 37 [33 to 41]
  4 Months: number analyzed (Participants) | 353 | 352
  4 Months | 40 [36 to 43] | 40 [36 to 43]
  12 Months: number analyzed (Participants) | 343 | 336
  12 Months | 41 [37 to 43] | 41 [38 to 45]
  24 Months: number analyzed (Participants) | 303 | 301
  24 Months | 41 [37 to 44] | 41 [37 to 44]
  36 Months: number analyzed (Participants) | 278 | 277
  36 Months | 40 [36 to 44] | 41 [38 to 45]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney) — 36 months

62. Secondary Outcome: H01: SF-12 Mental Component Summary (MCS) Scale
Description: Twelve items that reflect both physical and mental health are selected from the SF-36 subscales and combined according to an algebraic formula using published weights and constants: (a) First, the items are coded so that a higher value indicates better health; (b) then indicator variables (1/0) are created for the item response choice categories; (c) next, the 35 indicator variables are weighted using "mental" regression weights from the general US population and summed to produce the MCS-12 score; and (d) finally, a normalized score (with a mean of 50 and standard deviation of 10) is obtained by adding the "mental" constant from the scoring table to the sum of the 35 products.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 534 | 530
units on a scale
  Baseline | 44.6 (12.6) | 45.5 (13.0)
  4 Months: number analyzed (Participants) | 448 | 455
  4 Months | 50.5 (11.8) | 49.2 (12.3)
  12 Months: number analyzed (Participants) | 403 | 405
  12 Months | 51.8 (12.1) | 50.3 (12.6)
  24 Months: number analyzed (Participants) | 370 | 356
  24 Months | 51.6 (11.1) | 49.7 (12.6)
  36 Months: number analyzed (Participants) | 347 | 333
  36 Months | 51.6 (11.4) | 50.9 (11.9)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.004, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.011, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.007, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.044, Chi-squared — 36 months

63. Secondary Outcome: H02: SF-12 Mental Component Summary (MCS) Scale
Description: as for outcome 62
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 433 | 426
units on a scale
  Baseline | 42 [32 to 53] | 41 [33 to 53]
  4 Months: number analyzed (Participants) | 353 | 352
  4 Months | 54 [41 to 62] | 55 [44 to 61]
  12 Months: number analyzed (Participants) | 343 | 336
  12 Months | 57 [46 to 63] | 54 [45 to 62]
  24 Months: number analyzed (Participants) | 303 | 301
  24 Months | 56 [44 to 61] | 55 [44 to 62]
  36 Months: number analyzed (Participants) | 278 | 277
  36 Months | 56 [45 to 62] | 56 [46 to 62]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney) — 36 months

64. Secondary Outcome: H01: KCCQ Physical Limitation Scale
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ)Physical Limitation Scale: These 6 items assess ability to perform various activities of daily living. Response choices range from "Extremely limited" (1) to "Not at all limited" (5). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 597 | 585
units on a scale
  Baseline | 64.2 (24.7) | 64.7 (26.1)
  4 Months: number analyzed (Participants) | 511 | 527
  4 Months | 75.2 (23.6) | 73.1 (23.6)
  12 Months: number analyzed (Participants) | 472 | 464
  12 Months | 77.8 (23.0) | 73.4 (24.3)
  24 Months: number analyzed (Participants) | 410 | 412
  24 Months | 76.6 (23.1) | 73.1 (25.4)
  36 Months: number analyzed (Participants) | 404 | 385
  36 Months | 76.8 (22.0) | 74.9 (22.4)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.050, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.003, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority — 24 months; p = 0.049, Chi-squared
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.097, Chi-squared — 36 months

65. Secondary Outcome: H02: KCCQ Physical Limitation Scale
Description: These 6 items assess ability to perform various activities of daily living. Response choices range from "Extremely limited" (1) to "Not at all limited" (5). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 484 | 480
units on a scale
  Baseline | 63 [38 to 83] | 63 [45 to 80]
  4 Months: number analyzed (Participants) | 433 | 432
  4 Months | 83 [58 to 95] | 83 [64 to 96]
  12 Months: number analyzed (Participants) | 402 | 411
  12 Months | 84 [65 to 100] | 88 [67 to 96]
  24 Months: number analyzed (Participants) | 363 | 368
  24 Months | 88 [60 to 100] | 85 [66 to 96]
  36 Months: number analyzed (Participants) | 321 | 324
  36 Months | 88 [69 to 100] | 88 [67 to 96]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney) — 36 months

66. Secondary Outcome: H01: KCCQ Symptom Stability
Description: This item assesses changes in shortness of breath or fatigue over the past 2 weeks. Response choices range from "Much worse" (1) to "Much better" (5). Item score is transformed to a 0-100 scale with a high score representing a better outcome.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 604 | 590
units on a scale
  Baseline | 53.3 (23.3) | 55.5 (23.8)
  4 Months: number analyzed (Participants) | 513 | 534
  4 Months | 58.6 (20.5) | 55.7 (19.1)
  12 Months: number analyzed (Participants) | 470 | 470
  12 Months | 52.8 (15.7) | 51.1 (17.4)
  24 Months: number analyzed (Participants) | 413 | 415
  24 Months | 51.7 (14.5) | 49.3 (15.5)
  36 Months: number analyzed (Participants) | 411 | 390
  36 Months | 50.7 (14.4) | 50.8 (14.2)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.023, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney) — 36 months

67. Secondary Outcome: H02: KCCQ Symptom Stability
Description: This item assesses changes in shortness of breath or fatigue over the past 2 weeks. Response choices range from "Much worse" (1) to "Much better" (5). Item score is transformed to a 0-100 scale with a high score representing a better outcome.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 494 | 492
units on a scale
  Baseline | 50 [25 to 50] | 50 [50 to 50]
  4 Months: number analyzed (Participants) | 436 | 435
  4 Months | 50 [50 to 75] | 50 [50 to 75]
  12 Months: number analyzed (Participants) | 408 | 416
  12 Months | 50 [50 to 50] | 50 [50 to 50]
  24 Months: number analyzed (Participants) | 362 | 372
  24 Months | 50 [50 to 50] | 50 [50 to 50]
  36 Months: number analyzed (Participants) | 328 | 332
  36 Months | 50 [50 to 50] | 50 [50 to 50]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney) — 36 months

68. Secondary Outcome: H01: KCCQ Symptom Frequency
Description: These 4 items assess how many times the patient has been bothered by shortness of breath, fatigue, and ankle swelling over the past 2 weeks. Response choices vary, but they range from "Every morning" or "Every night" or "All of the time" (1) to "Never over the past 2 weeks" (either 5 or 7). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 606 | 592
units on a scale
  Baseline | 70.5 (24.6) | 71.5 (25.7)
  4 Months: number analyzed (Participants) | 519 | 534
  4 Months | 79.8 (21.6) | 79.1 (21.8)
  12 Months: number analyzed (Participants) | 475 | 471
  12 Months | 82.4 (22.2) | 79.2 (23.5)
  24 Months: number analyzed (Participants) | 415 | 417
  24 Months | 82.2 (20.9) | 79.3 (23.3)
  36 Months: number analyzed (Participants) | 411 | 391
  36 Months | 81.7 (22.7) | 80.4 (22.4)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.205, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.017, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG; Test type: Superiority; p = 0.028, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.123, Chi-squared — 36 months

69. Secondary Outcome: H02: KCCQ Symptom Frequency
Description: These 4 items assess how many times the patient has been bothered by shortness of breath, fatigue, and ankle swelling over the past 2 weeks. Response choices vary, but they range from "Every morning" or "Every night" or "All of the time" (1) to "Never over the past 2 weeks" (either 5 or 7). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 493 | 491
units on a scale
  Baseline | 67 [50 to 88] | 71 [50 to 88]
  4 Months: number analyzed (Participants) | 440 | 434
  4 Months | 83 [63 to 100] | 88 [67 to 100]
  12 Months: number analyzed (Participants) | 409 | 415
  12 Months | 90 [67 to 100] | 90 [71 to 100]
  24 Months: number analyzed (Participants) | 367 | 374
  24 Months | 92 [67 to 100] | 92 [69 to 100]
  36 Months: number analyzed (Participants) | 329 | 334
  36 Months | 92 [67 to 100] | 92 [69 to 100]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney) — 36 months

70. Secondary Outcome: H01: KCCQ Symptom Burden
Description: These 3 items assess how much the patient has been bothered by shortness of breath, fatigue, and ankle swelling over the past 2 weeks. Response choices range from "extremely bothersome" (1) to "Not at all bothersome" (5). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 606 | 591
units on a scale
  Baseline | 72.6 (22.5) | 73.4 (24.4)
  4 Months: number analyzed (Participants) | 517 | 535
  4 Months | 81.4 (20.4) | 79.6 (21.0)
  12 Months: number analyzed (Participants) | 475 | 471
  12 Months | 83.7 (20.6) | 79.8 (22.5)
  24 Months: number analyzed (Participants) | 415 | 417
  24 Months | 83.3 (20.2) | 80.0 (23.1)
  36 Months: number analyzed (Participants) | 411 | 391
  36 Months | 83.1 (21.2) | 80.7 (22.4)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.050, Chi-squared — 4 months; P-values were based on the Chi-Square test applied to maximum likelihood estimates derived from an adjusted mixed model
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.006, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.039, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.074, Chi-squared — 36 months

71. Secondary Outcome: H02: KCCQ Symptom Burden
Description: as for outcome 70
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 494 | 492
units on a scale
  Baseline | 67 [50 to 92] | 75 [50 to 83]
  4 Months: number analyzed (Participants) | 441 | 436
  4 Months | 83 [67 to 100] | 83 [67 to 100]
  12 Months: number analyzed (Participants) | 410 | 416
  12 Months | 92 [67 to 100] | 92 [67 to 100]
  24 Months: number analyzed (Participants) | 368 | 373
  24 Months | 92 [67 to 100] | 92 [67 to 100]
  36 Months: number analyzed (Participants) | 329 | 332
  36 Months | 92 [67 to 100] | 92 [67 to 100]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.35, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney) — 36 months

72. Secondary Outcome: H01: KCCQ Total Symptoms
Description: This score represents the mean of the Symptom Frequency and Symptom Burden scores. Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 606 | 592
units on a scale
  Baseline | 71.7 (22.5) | 72.6 (24.2)
  4 Months: number analyzed (Participants) | 519 | 535
  4 Months | 80.8 (20.0) | 79.5 (20.5)
  12 Months: number analyzed (Participants) | 475 | 471
  12 Months | 83.2 (20.5) | 79.6 (22.1)
  24 Months: number analyzed (Participants) | 415 | 417
  24 Months | 82.9 (19.8) | 79.8 (22.6)
  36 Months: number analyzed (Participants) | 411 | 391
  36 Months | 82.5 (21.3) | 80.7 (21.7)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.085, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.007, Chi-squared
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.026, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.085, Chi-squared — 36 months

73. Secondary Outcome: H02: KCCQ Total Symptoms
Description: This score represents the mean of the Symptom Frequency and Symptom Burden scores. Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 494 | 492
units on a scale
  Baseline | 68 [48 to 86] | 71 [52 to 88]
  4 Months: number analyzed (Participants) | 441 | 436
  4 Months | 84 [65 to 100] | 88 [71 to 100]
  12 Months: number analyzed (Participants) | 410 | 416
  12 Months | 90 [68 to 100] | 88 [71 to 100]
  24 Months: number analyzed (Participants) | 368 | 374
  24 Months | 90 [71 to 100] | 90 [71 to 100]
  36 Months: number analyzed (Participants) | 329 | 334
  36 Months | 90 [70 to 100] | 92 [68 to 100]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney) — 36 months

74. Secondary Outcome: H01: KCCQ Quality-of-Life Scale
Description: These 3 items assess the effect of heart failure on the patient's enjoyment of life. Response choices range from 1 (worst state) to 5 (best state). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 606 | 591
units on a scale
  Baseline | 47.9 (25.0) | 50.1 (27.0)
  4 Months: number analyzed (Participants) | 519 | 533
  4 Months | 68.7 (24.5) | 63.3 (25.6)
  12 Months: number analyzed (Participants) | 472 | 469
  12 Months | 72.9 (23.5) | 65.6 (25.8)
  24 Months: number analyzed (Participants) | 416 | 417
  24 Months | 71.9 (22.6) | 66.9 (26.0)
  36 Months: number analyzed (Participants) | 410 | 390
  36 Months | 71.2 (23.3) | 69.1 (24.8)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 12 month
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.018, Chi-squared — 36 months

75. Secondary Outcome: H02: KCCQ Quality-of-Life Scale
Description: These 3 items assess the effect of heart failure on the patient's enjoyment of life. Response choices range from 1 (worst state) to 5 (best state). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 493 | 490
units on a scale
  Baseline | 42 [17 to 58] | 33 [25 to 58]
  4 Months: number analyzed (Participants) | 441 | 433
  4 Months | 75 [50 to 92] | 75 [58 to 92]
  12 Months: number analyzed (Participants) | 409 | 416
  12 Months | 75 [50 to 92] | 75 [58 to 92]
  24 Months: number analyzed (Participants) | 365 | 373
  24 Months | 75 [58 to 92] | 75 [58 to 92]
  36 Months: number analyzed (Participants) | 328 | 333
  36 Months | 75 [58 to 92] | 83 [58 to 92]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.70, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.84, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney) — 36 months

76. Secondary Outcome: H01: KCCQ Social Limitation
Description: These 4 items assess how much heart failure has affected the patient's lifestyle. Response choices range from "Severely limited" (1) to "Did not limit at all" (5). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 570 | 554
units on a scale
  Baseline | 56.4 (29.9) | 57.3 (29.7)
  4 Months: number analyzed (Participants) | 495 | 510
  4 Months | 72.3 (27.4) | 69.0 (27.0)
  12 Months: number analyzed (Participants) | 453 | 445
  12 Months | 76.4 (26.0) | 69.5 (28.4)
  24 Months: number analyzed (Participants) | 395 | 402
  24 Months | 75.4 (25.9) | 71.0 (28.8)
  36 Months: number analyzed (Participants) | 399 | 374
  36 Months | 75.4 (27.0) | 72.8 (26.8)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.023, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.001, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.077, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.170, Chi-squared — 36 months

77. Secondary Outcome: H02: KCCQ Social Limitation
Description: These 4 items assess how much heart failure has affected the patient's lifestyle. Response choices range from "Severely limited" (1) to "Did not limit at all" (5). Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 465 | 467
units on a scale
  Baseline | 44 [19 to 75] | 44 [25 to 75]
  4 Months: number analyzed (Participants) | 424 | 412
  4 Months | 75 [50 to 94] | 75 [50 to 100]
  12 Months: number analyzed (Participants) | 387 | 400
  12 Months | 81 [58 to 100] | 83 [63 to 94]
  24 Months: number analyzed (Participants) | 353 | 356
  24 Months | 81 [50 to 100] | 86 [56 to 100]
  36 Months: number analyzed (Participants) | 318 | 309
  36 Months | 83 [58 to 100] | 83 [56 to 100]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — 36 months

78. Secondary Outcome: H01: KCCQ Clinical Summary Score
Description: This score represents the mean of the Physical Limitation and Total Symptom scores. Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 607 | 592
units on a scale
  Baseline | 68.2 (21.8) | 68.8 (23.1)
  4 Months: number analyzed (Participants) | 520 | 537
  4 Months | 78.2 (20.0) | 76.4 (20.4)
  12 Months: number analyzed (Participants) | 476 | 473
  12 Months | 80.6 (20.3) | 76.4 (21.9)
  24 Months: number analyzed (Participants) | 418 | 417
  24 Months | 80.1 (19.5) | 76.6 (22.6)
  36 Months: number analyzed (Participants) | 412 | 391
  36 Months | 79.9 (20.2) | 78.0 (20.5)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.033, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.002, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.015, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.051, Chi-squared — 36 months

79. Secondary Outcome: H02: KCCQ Clinical Summary Score
Description: This score represents the mean of the Physical Limitation and Total Symptom scores. Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 496 | 492
units on a scale
  Baseline | 65 [46 to 83] | 68 [49 to 84]
  4 Months: number analyzed (Participants) | 445 | 443
  4 Months | 84 [63 to 95] | 84 [67 to 96]
  12 Months: number analyzed (Participants) | 411 | 416
  12 Months | 88 [66 to 97] | 86 [70 to 96]
  24 Months: number analyzed (Participants) | 368 | 374
  24 Months | 88 [65 to 97] | 87 [69 to 96]
  36 Months: number analyzed (Participants) | 329 | 335
  36 Months | 88 [67 to 98] | 88 [69 to 98]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney) — 36 months

80. Secondary Outcome: H01: KCCQ Overall Summary Score
Description: This score represents the mean of these 4 scores: Physical Limitation, Total Symptom, Quality of Life, and Social Limitation. Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 607 | 592
units on a scale
  Baseline | 60.3 (22.3) | 61.3 (23.2)
  4 Months: number analyzed (Participants) | 520 | 537
  4 Months | 74.3 (21.0) | 71.2 (21.3)
  12 Months: number analyzed (Participants) | 476 | 473
  12 Months | 77.5 (20.4) | 72.2 (22.7)
  24 Months: number analyzed (Participants) | 418 | 417
  24 Months | 76.9 (20.1) | 72.9 (23.4)
  36 Months: number analyzed (Participants) | 412 | 391
  36 Months | 76.6 (20.9) | 74.5 (21.4)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.006, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.037, Chi-squared — 36 months

81. Secondary Outcome: H02: KCCQ Overall Summary Score
Description: This score represents the mean of these 4 scores: Physical Limitation, Total Symptom, Quality of Life, and Social Limitation. Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 496 | 492
units on a scale
  Baseline | 53 [36 to 70] | 54 [38 to 72]
  4 Months: number analyzed (Participants) | 446 | 443
  4 Months | 79 [56 to 92] | 79 [63 to 92]
  12 Months: number analyzed (Participants) | 411 | 416
  12 Months | 84 [59 to 95] | 82 [66 to 94]
  24 Months: number analyzed (Participants) | 368 | 374
  24 Months | 84 [60 to 95] | 84 [64 to 94]
  36 Months: number analyzed (Participants) | 329 | 335
  36 Months | 85 [65 to 95] | 84 [63 to 95]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney) — 36 months

82. Secondary Outcome: H01: Seattle Angina Questionnaire (SAQ) Anginal Frequency Subscale
Description: These 2 items assess the frequency of chest pain over the last 4 weeks. Response choices range from "4 or more times a day" (1) to "None" (6). The mean response is transformed to a 0-100 scale where higher scores reflect less frequent angina.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 594 | 584
units on a scale
  Baseline | 74.3 (26.7) | 77.0 (26.2)
  4 Months: number analyzed (Participants) | 506 | 522
  4 Months | 90.5 (16.9) | 84.0 (23.2)
  12 Months: number analyzed (Participants) | 459 | 458
  12 Months | 90.6 (16.5) | 84.0 (22.4)
  24 Months: number analyzed (Participants) | 404 | 403
  24 Months | 90.5 (17.2) | 86.5 (19.7)
  36 Months: number analyzed (Participants) | 395 | 372
  36 Months | 89.8 (17.5) | 88.5 (19.0)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.010, Chi-squared — 36 months

83. Secondary Outcome: H02: Seattle Angina Questionnaire (SAQ) Anginal Frequency Subscale
Description: These 2 items assess the frequency of chest pain over the last 4 weeks. Response choices range from "4 or more times a day" (1) to "None" (6). The mean response is transformed to a 0-100 scale where higher scores reflect less frequent angina.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 488 | 482
units on a scale
  Baseline | 70 [40 to 90] | 80 [50 to 100]
  4 Months: number analyzed (Participants) | 414 | 412
  4 Months | 100 [90 to 100] | 100 [90 to 100]
  12 Months: number analyzed (Participants) | 379 | 392
  12 Months | 100 [90 to 100] | 100 [90 to 100]
  24 Months: number analyzed (Participants) | 345 | 351
  24 Months | 100 [80 to 100] | 100 [90 to 100]
  36 Months: number analyzed (Participants) | 310 | 314
  36 Months | 100 [90 to 100] | 100 [90 to 100]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney) — 36 months

84. Secondary Outcome: H01: Seattle Angina Questionnaire (SAQ) Anginal Stability Subscale
Description: This item assesses the change in chest pain over the last 4 weeks. Response choices range from "Much more often" (1) to "None" (6). The mean response is transformed to a 0-100 scale where 50 represents no change and a higher score indicates less angina.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 575 | 565
units on a scale
  Baseline | 56.0 (27.1) | 57.8 (25.0)
  4 Months: number analyzed (Participants) | 503 | 515
  4 Months | 58.3 (20.3) | 55.8 (20.6)
  12 Months: number analyzed (Participants) | 459 | 456
  12 Months | 55.4 (17.3) | 53.3 (17.6)
  24 Months: number analyzed (Participants) | 402 | 402
  24 Months | 52.9 (14.9) | 52.9 (17.4)
  36 Months: number analyzed (Participants) | 394 | 366
  36 Months | 53.9 (16.9) | 53.6 (15.5)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.029, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.042, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.30, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.20, Chi-squared — 36 months

85. Secondary Outcome: H02: Seattle Angina Questionnaire (SAQ) Anginal Stability Subscale
Description: This item assesses the change in chest pain over the last 4 weeks. Response choices range from "Much more often" (1) to "None" (6). The mean response is transformed to a 0-100 scale where 50 represents no change and a higher score indicates less angina.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 477 | 462
units on a scale
  Baseline | 50 [25 to 50] | 50 [25 to 50]
  4 Months: number analyzed (Participants) | 411 | 405
  4 Months | 50 [50 to 50] | 50 [50 to 50]
  12 Months: number analyzed (Participants) | 374 | 388
  12 Months | 50 [50 to 50] | 50 [50 to 50]
  24 Months: number analyzed (Participants) | 344 | 349
  24 Months | 50 [50 to 50] | 50 [50 to 50]
  36 Months: number analyzed (Participants) | 310 | 313
  36 Months | 50 [50 to 50] | 50 [50 to 50]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney) — 36 months

86. Secondary Outcome: H01:Seattle Angina Questionnaire (SAQ) Quality-of-Life Subscale
Description: These 3 items measure the patient's general satisfaction with life. Response choices range from 1 (least enjoyment) to 5 (high satisfaction). The mean score is transformed to a 0-100 scale where higher scores reflect better outcomes.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 585 | 574
units on a scale
  Baseline | 53.6 (25.9) | 57.6 (26.6)
  4 Months: number analyzed (Participants) | 505 | 525
  4 Months | 74.5 (22.1) | 67.5 (24.4)
  12 Months: number analyzed (Participants) | 457 | 457
  12 Months | 75.8 (21.2) | 69.1 (24.0)
  24 Months: number analyzed (Participants) | 401 | 404
  24 Months | 75.5 (21.5) | 68.7 (24.9)
  36 Months: number analyzed (Participants) | 395 | 371
  36 Months | 75.3 (22.1) | 72.9 (22.2)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.001, Chi-squared — 36 months

87. Secondary Outcome: H02: Seattle Angina Questionnaire (SAQ) Quality-of-Life Subscale
Description: These 3 items measure the patient's general satisfaction with life. Response choices range from 1 (least enjoyment) to 5 (high satisfaction). The mean score is transformed to a 0-100 scale where higher scores reflect better outcomes.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 484 | 478
units on a scale
  Baseline | 42 [25 to 67] | 42 [25 to 67]
  4 Months | 83 [67 to 100] | 83 [58 to 92]
  12 Months | 83 [67 to 100] | 83 [67 to 100]
  24 Months | 83 [58 to 100] | 83 [67 to 100]
  36 Months | 83 [67 to 100] | 83 [67 to 100]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — 36 months

88. Secondary Outcome: H01: EQ-5D Visual Analog Scale
Description: Euro QoL 5 Dimensions Quality of Life Instrument (EQ-5D): This 0-100 scale records the patient's self-rated health on a vertical scale where 0 = worst imaginable health and 100 = perfect health.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 593 | 585
units on a scale
  Baseline | 56.7 (19.0) | 59.5 (18.8)
  4 Months: number analyzed (Participants) | 497 | 518
  4 Months | 68.5 (18.1) | 65.4 (17.7)
  12 Months: number analyzed (Participants) | 447 | 455
  12 Months | 69.2 (17.9) | 65.4 (18.5)
  24 Months: number analyzed (Participants) | 390 | 398
  24 Months | 68.6 (17.8) | 65.9 (18.4)
  36 Months: number analyzed (Participants) | 384 | 378
  36 Months | 69.0 (17.9) | 67.1 (17.4)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.001, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.001, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.001, Chi-squared

89. Secondary Outcome: H02: EQ-5D Visual Analog Scale
Description: This 0-100 scale records the patient's self-rated health on a vertical scale where 0 = worst imaginable health and 100 = perfect health.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 488 | 487
units on a scale
  Baseline | 50 [40 to 70] | 50 [40 to 70]
  4 Months: number analyzed (Participants) | 420 | 415
  4 Months | 70 [60 to 80] | 70 [60 to 80]
  12 Months: number analyzed (Participants) | 383 | 385
  12 Months | 72 [60 to 80] | 70 [60 to 80]
  24 Months: number analyzed (Participants) | 371 | 352
  24 Months | 70 [50 to 80] | 70 [50 to 80]
  36 Months: number analyzed (Participants) | 330 | 331
  36 Months | 70 [50 to 80] | 70 [52 to 80]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney) — 36 months

90. Secondary Outcome: H01: EQ-5D Health Status Index Score
Description: This 5-item scale describes a patient's health in terms of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Choices for each dimension are "No problems" (1), "Moderate problems" (2), or "Extreme problems" (3). A scoring algorithm with utility weights is then applied to these 5 items to generate index scores ranging from -0.11 (i.e., 33333) to 1.0 (i.e., 11111) on a scale where 0.0 = death and 1.0 = perfect health. These scores were multiplied by 100 to produce a scale from -11 to 100 that more closely resembles the Visual Analog Scale.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 584 | 570
units on a scale
  Baseline | 69.3 (25.8) | 72.3 (24.4)
  4 Months: number analyzed (Participants) | 489 | 504
  4 Months | 78.9 (24.5) | 77.4 (22.6)
  12 Months: number analyzed (Participants) | 439 | 453
  12 Months | 80.5 (22.3) | 77.6 (24.0)
  24 Months: number analyzed (Participants) | 386 | 394
  24 Months | 79.6 (24.6) | 78.1 (25.9)
  36 Months: number analyzed (Participants) | 379 | 371
  36 Months | 81.4 (23.4) | 81.5 (21.6)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.007, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.003, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.023, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.060, Chi-squared — 36 months

91. Secondary Outcome: H02: EQ-5D Health Status Index Score
Description: This 5-item scale describes a patient's health in terms of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Choices for each dimension are "No problems" (1), "Moderate problems" (2), or "Extreme problems" (3). A scoring algorithm with utility weights is then applied to these 5 items to generate index scores ranging from -0.11 (i.e., 33333) to 1.0 (i.e., 11111) on a scale where 0.0 = death and 1.0 = perfect health. (These scores can be multiplied by 100 to produce a scale from -11 to 100 that more closely resembles the Visual Analog Scale.)
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 475 | 477
units on a scale
  Baseline | 69 [52 to 81] | 69 [59 to 81]
  4 Months: number analyzed (Participants) | 405 | 395
  4 Months | 85 [69 to 100] | 85 [69 to 100]
  12 Months: number analyzed (Participants) | 375 | 379
  12 Months | 85 [73 to 100] | 85 [73 to 100]
  24 Months: number analyzed (Participants) | 356 | 339
  24 Months | 85 [69 to 100] | 85 [69 to 100]
  36 Months: number analyzed (Participants) | 323 | 322
  36 Months | 85 [69 to 100] | 85 [69 to 100]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney) — 36 months

92. Secondary Outcome: H01: Percentage of Patients With a Score of >= 16 on the Center for Epidemiological Studies Depression (CES-D) Scale
Description: These 20 items assess depressive symptomatology, and responses choices range from "Rarely or none of the time" (0) to "Most or all of the time" (3). Scale scores can therefore range from 0 to 60, although scores greater than or equal to 16 are considered high.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 595 | 583
percentage of participants
  Baseline | 42.9 | 43.4
  4 Months: number analyzed (Participants) | 501 | 521
  4 Months | 26.6 | 27.5
  12 Months: number analyzed (Participants) | 457 | 454
  12 Months | 25.0 | 26.9
  24 Months: number analyzed (Participants) | 399 | 402
  24 Months | 24.1 | 31.1
  36 Months: number analyzed (Participants) | 393 | 370
  36 Months | 22.4 | 29.5
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.86, Chi-squared — Baseline; All P-values were based on the Likelihood Ratio Chi-Square test
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.78, Chi-squared — 4 months; All P-values were based on the Likelihood Ratio Chi-Square test
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.55, Chi-squared — 12 months; All P-values were based on the Likelihood Ratio Chi-Square test
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.027, Chi-squared — 24 months; All P-values were based on the Likelihood Ratio Chi-Square test
Statistical Analysis 5: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.031, Chi-squared — 36 months; All P-values were based on the Likelihood Ratio Chi-Square test

93. Secondary Outcome: H02: Percentage of Patients With a Score of >= 16 on the Center for Epidemiological Studies Depression (CES-D) Scale
Description: These 20 items assess depressive symptomatology, and responses choices range from "Rarely or none of the time" (0) to "Most or all of the time" (3). Scale scores can therefore range from 0 to 60, although scores greater than or equal to 16 are considered high.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 496 | 495
percentage of participants
  Baseline | 50.5 | 53.2
  4 Months: number analyzed (Participants) | 449 | 448
  4 Months | 29.6 | 27.0
  12 Months: number analyzed (Participants) | 411 | 417
  12 Months | 24.4 | 27.0
  24 Months: number analyzed (Participants) | 371 | 379
  24 Months | 28.1 | 24.3
  36 Months: number analyzed (Participants) | 333 | 336
  36 Months | 20.8 | 24.8
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.40, Chi-squared — Baseline; All P-values were based on the Likelihood Ratio Chi-Square test
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.42, Chi-squared — 4 months; All P-values were based on the Likelihood Ratio Chi-Square test
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.41, Chi-squared — 12 months; All P-values were based on the Likelihood Ratio Chi-Square test
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.25, Chi-squared — 24 months; All P-values were based on the Likelihood Ratio Chi-Square test
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.25, Chi-squared — 36 months; All P-values were based on the Likelihood Ratio Chi-Square test

94. Secondary Outcome: H01: Cardiac Self-Efficacy (CSE) Maintain Functioning Subscale
Description: These 5 items assess patients' ability to maintain their usual social, family, and physical activities. Response choices range from "Not at all confident" (1) to "Completely confident" (5). The mean score is transformed to a 0-100 scale where higher scores reflect more confidence.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 596 | 581
units on a scale
  Baseline | 46.8 (24.3) | 49.3 (24.9)
  4 Months: number analyzed (Participants) | 504 | 521
  4 Months | 56.0 (25.0) | 53.8 (24.8)
  12 Months: number analyzed (Participants) | 455 | 456
  12 Months | 56.7 (25.9) | 53.9 (26.7)
  24 Months: number analyzed (Participants) | 399 | 401
  24 Months | 55.3 (25.2) | 53.3 (26.4)
  36 Months: number analyzed (Participants) | 392 | 370
  36 Months | 56.2 (26.0) | 54.9 (26.7)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.002, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.007, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.049, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.038, Chi-squared — 36 months

95. Secondary Outcome: H02: Cardiac Self-Efficacy (CSE) Maintain Functioning Subscale
Description: These 5 items assess patients' ability to maintain their usual social, family, and physical activities. Response choices range from "Not at all confident" (1) to "Completely confident" (5). The mean score is transformed to a 0-100 scale where higher scores reflect more confidence.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 487 | 481
units on a scale
  Baseline | 45 [25 to 63] | 45 [25 to 67]
  4 Months: number analyzed (Participants) | 406 | 409
  4 Months | 61 [38 to 75] | 63 [40 to 75]
  12 Months: number analyzed (Participants) | 381 | 386
  12 Months | 65 [42 to 80] | 64 [45 to 75]
  24 Months: number analyzed (Participants) | 344 | 347
  24 Months | 63 [44 to 78] | 65 [45 to 80]
  36 Months: number analyzed (Participants) | 306 | 307
  36 Months | 58 [40 to 75] | 63 [45 to 75]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney) — 36 months

96. Secondary Outcome: H01: Cardiac Self-Efficacy (CSE) Control Symptoms Subscale
Description: These 8 items assess patients' ability to control symptoms such as chest pain and breathlessness by taking their medications and adjusting their activity levels. Response choices range from "Not at all confident" (1) to "Completely confident" (5). The mean score is transformed to a 0-100 scale where higher scores reflect more confidence.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 599 | 583
units on a scale
  Baseline | 62.9 (22.5) | 64.8 (21.2)
  4 Months: number analyzed (Participants) | 504 | 522
  4 Months | 69.2 (20.6) | 68.7 (20.5)
  12 Months: number analyzed (Participants) | 454 | 458
  12 Months | 68.7 (20.3) | 67.4 (21.8)
  24 Months: number analyzed (Participants) | 401 | 403
  24 Months | 68.3 (20.4) | 66.2 (21.3)
  36 Months: number analyzed (Participants) | 393 | 370
  36 Months | 69.7 (21.0) | 68.3 (21.1)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.036, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.043, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.018, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.037, Chi-squared — 36 months

97. Secondary Outcome: H02: Cardiac Self-Efficacy (CSE) Control Symptoms Subscale
Description: These 8 items assess patients' ability to control symptoms such as chest pain and breathlessness by taking their medications and adjusting their activity levels. Response choices range from "Not at all confident" (1) to "Completely confident" (5). The mean score is transformed to a 0-100 scale where higher scores reflect more confidence.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 487 | 482
units on a scale
  Baseline | 63 [47 to 75] | 63 [47 to 75]
  4 Months: number analyzed (Participants) | 412 | 409
  4 Months | 75 [62 to 91] | 75 [61 to 88]
  12 Months: number analyzed (Participants) | 381 | 387
  12 Months | 75 [63 to 91] | 75 [63 to 88]
  24 Months: number analyzed (Participants) | 346 | 347
  24 Months | 75 [63 to 92] | 75 [61 to 88]
  36 Months: number analyzed (Participants) | 311 | 314
  36 Months | 75 [63 to 84] | 75 [63 to 91]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.75, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — 36 months

98. Secondary Outcome: H01: General Health Rating Scale
Description: This single item asks patients to describe their health status over the past month on a scale from 0 to 100, where 0 = death and 100 = excellent health.
  .
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 579 | 554
units on a scale
  Baseline | 56.0 (19.4) | 57.6 (19.0)
  4 Months: number analyzed (Participants) | 486 | 493
  4 Months | 67.3 (19.1) | 64.0 (18.1)
  12 Months: number analyzed (Participants) | 438 | 437
  12 Months | 68.7 (18.7) | 63.7 (19.1)
  24 Months: number analyzed (Participants) | 388 | 391
  24 Months | 68.1 (19.2) | 65.0 (19.6)
  36 Months: number analyzed (Participants) | 385 | 364
  36 Months | 69.1 (31.6) | 67.1 (33.7)
Statistical Analysis 1: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.0002, Chi-squared — 4 months; [statistical method as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.0001, Chi-squared — 12 months
Statistical Analysis 3: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.009, Chi-squared — 24 months
Statistical Analysis 4: Comparison: Total H01: Medication + CABG vs H01: Medication; Test type: Superiority; p = 0.32, Chi-squared — 36 months

99. Secondary Outcome: H02: General Health Rating Scale
Description: This single item asks patients to describe their health status over the past month on a scale from 0 to 100, where 0 = death and 100 = excellent health.
Time Frame: From enrollment to 3-year follow-up
Population: Only patients with questionnaire data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 466 | 458
units on a scale
  Baseline | 50 [40 to 70] | 50 [40 to 70]
  4 Months: number analyzed (Participants) | 387 | 389
  4 Months | 70 [50 to 80] | 70 [60 to 80]
  12 Months: number analyzed (Participants) | 367 | 370
  12 Months | 70 [50 to 80] | 70 [60 to 80]
  24 Months: number analyzed (Participants) | 338 | 339
  24 Months | 70 [50 to 80] | 70 [50 to 80]
  36 Months: number analyzed (Participants) | 298 | 303
  36 Months | 70 [60 to 80] | 70 [55 to 80]
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney) — Baseline
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.14, Wilcoxon (Mann-Whitney) — 4 months
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney) — 12 months
Statistical Analysis 4: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney) — 24 months
Statistical Analysis 5: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.84, Wilcoxon (Mann-Whitney) — 36 months

100. Secondary Outcome: H01: Cost of Care
Description: Hospital costs and physician fees for US patients
Time Frame: index hospital admission
Population: US patients with hospital bills
Measure: Mean (Standard Deviation); unit: 2009 US Dollars
Groups:
- H01: Medication + CABG: Coronary artery bypass graft surgery (CABG) plus Medication to treat coronary artery disease
  CABG surgery plus MED (medication): CABG plus standard medication management for Coronary Artery Disease
Arm/Group | H01: Medication + CABG | H01: Medication
Number analyzed (Participants) | 66 | 54
2009 US Dollars
  Hospital Costs | 50,032 (41,622) | 8,315 (19,719)
  Physician Fees | 5,405 (2,377) | 408 (819)
  Total Index Cost | 55,437 (43,460) | 8,723 (20,506)
Statistical Analysis 1: Comparison: H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — Hospital costs
Statistical Analysis 2: Comparison: H01: Medication + CABG; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — Physician fees
Statistical Analysis 3: Comparison: H01: Medication + CABG vs H01: Medication; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — Total index cost

101. Secondary Outcome: H02: Cost of Care
Description: Hospital costs and physician fees for US patients
Time Frame: index hospital admission
Population: US patients with hospital bills
Measure: Mean (Standard Deviation); unit: 2008 US Dollars
Arm/Group | H02: Medication+CABG | H02: Medication+CABG+SVR
Number analyzed (Participants) | 100 | 96
2008 US Dollars
  Hospital Costs | 50,939 (46,458) | 64,202 (49,172)
  Physician Fees | 5,183 (2,306) | 6,515 (2,463)
  Total Index Cost | 56,122 (48,552) | 70,717 (51,367)
Statistical Analysis 1: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney) — Hospital costs
Statistical Analysis 2: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — Physician fees
Statistical Analysis 3: Comparison: H02: Medication+CABG vs H02: Medication+CABG+SVR; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney) — Total index cost

ADVERSE EVENTS:
Time Frame: No "other" adverse events were collected, however serious adverse events were collected for the first 5 years of the follow up period per study protocol.
Arm/Group | H01: Medication | H01: Medication + CABG | H01 & H02: Medication+CABG | H02: Medication+CABG | H02: Medication+CABG+SVR
Serious Adverse Events (participants affected / at risk) | 84/602 | 85/534 | 9/76 | 31/423 | 53/501
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | H01: Medication (N=602) | H01: Medication + CABG (N=534) | H01 & H02: Medication+CABG (N=76) | H02: Medication+CABG (N=423) | H02: Medication+CABG+SVR (N=501)
ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
ACUTE HEART FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 4 | 0 | 0 | 0
ACUTE PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
ACUTE RENAL FAILURE (Renal and urinary disorders) | 0 | 7 | 1 | 4 | 9
ACUTE RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
ALS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
ANGINAL DISCOMFORT (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
ANOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
AORTIC RUPTURE (Vascular disorders) | 0 | 0 | 0 | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 6 | 7 | 0 | 1 | 4
ARTERIAL EMBOLISM (LIMBS) (Vascular disorders) | 4 | 3 | 0 | 0 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ASPIRATION PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
ASYSTOLIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1 | 0 | 2 | 0
BACTEREMIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
BOWEL ISCHEMIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
BRAIN TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
BUN INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
CANCER OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 5 | 5 | 0 | 0 | 2
CARDIAC ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
CARDIAC CIRRHOSIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
CARDIAC DISORDER (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
CARDIAC FAILURE AGGRAVATED (Cardiac disorders) | 2 | 0 | 0 | 1 | 1
CARDIAC TAMPONADE (Cardiac disorders) | 1 | 1 | 0 | 0 | 1
CARDIAC VENTRICULAR THROMBOSIS (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 3 | 3 | 0 | 2 | 2
CARDIOPULMONARY INSUFFICIENCY (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
CHRONIC SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
CLAUDICATION (Vascular disorders) | 1 | 0 | 0 | 0 | 0
CMV INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
CONFUSION (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
CONGESTIVE CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
CONGESTIVE HEART FAILURE (Cardiac disorders) | 3 | 2 | 0 | 0 | 1
CORONARY OCCLUSION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CREATININE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
CYSTITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
DECOMPENSATED HEART FAILURE (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
DECOMPENSATION CARDIAC (Cardiac disorders) | 0 | 1 | 0 | 0 | 2
DEVICE LEAD ISSUE (General disorders) | 1 | 0 | 0 | 0 | 0
DIARRHEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
EDEMA (General disorders) | 0 | 0 | 0 | 0 | 1
EDEMA PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
EMBOLIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
END STAGE CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
GALLSTONES (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
GASTRIC ULCER PERFORATED (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
GOUT (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 | 0 | 0 | 0 | 1
HEART FAILURE (Cardiac disorders) | 11 | 6 | 1 | 3 | 2
HEMODYNAMIC INSTABILITY (Vascular disorders) | 1 | 0 | 0 | 0 | 0
HEMORRHAGE BRAIN (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
HEPATIC INSUFFICIENCY (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
HEPATOMEGALY (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
HERNIA (General disorders) | 0 | 1 | 0 | 0 | 0
HOSPITALIZATION NOS (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 1 | 0
HYPOVOLEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
IMPLANT SITE INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
INFECTED SKIN ULCER (Infections and infestations) | 0 | 0 | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 2
INSUFFICIENCY CARDIAC (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
ISCHEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
LOW BLOOD PRESSURE (Vascular disorders) | 2 | 0 | 0 | 0 | 0
LOW CARDIAC OUTPUT SYNDROME (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
MALIGNANT VENTRICULAR ARRHYTHMIAS (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
MEDIASTINAL HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
MEDIASTINITIS (Infections and infestations) | 0 | 4 | 0 | 0 | 0
MESOTHELIOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
MITRAL VALVE DISEASE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
MULTI ORGAN FAILURE (General disorders) | 0 | 1 | 0 | 0 | 0
MULTIORGAN FAILURE (General disorders) | 0 | 0 | 0 | 0 | 1
MULTIPLE ORGAN FAILURE (General disorders) | 0 | 0 | 1 | 0 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 3 | 0 | 2 | 2
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
NECROSIS SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
NECROTIZING FASCIITIS (Infections and infestations) | 1 | 1 | 0 | 0 | 0
OTHER CARDIAC (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
PAROXYSMAL ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
PERIPHERAL VASCULAR DISEASE (Vascular disorders) | 0 | 1 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 2
PNEUMONIA (Infections and infestations) | 1 | 1 | 0 | 0 | 1
POSTOPERATIVE HEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
POSTPERICARDIOTOMY SYNDROME (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
PULMONARY EMBOLUS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
PULMONARY THROMBOEMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
RENAL INSUFFICIENCY (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
SCLERODERMA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
SEPSIS (Infections and infestations) | 1 | 1 | 0 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 1 | 0 | 0 | 1
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
SIRS (General disorders) | 0 | 0 | 0 | 0 | 1
SKIN TROPHIC ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
STERNAL DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
STROKE (Nervous system disorders) | 17 | 16 | 2 | 9 | 10
SUPERFICIAL PHLEBOTHROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0
SUSTAINED VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
SVT (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
UNSTABLE ANGINA (Cardiac disorders) | 2 | 0 | 0 | 0 | 1
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 2 | 4 | 0 | 1 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 6 | 3 | 2 | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 2
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
VOLUME OVERLOAD (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement is that all publications need to be reviewed and approved by the Policy and Publication Committee and the Sponsor prior to publication.